

| Document Title: | Statistical Analysis Plan BIO Master.Cor Family |
|---|---|
| Document Version and Date: | Version 3-0, 18-Mar-2022 |
| ClinicalTrials.gov Identifier: | NCT03891329 |

# Cover Sheet Statistical Analysis Plan BIO|Master.Cor Family Version 3-0

FOR-137-059 Rev. B

Page 1/88

| Sponsor: | Biotronik SE & Co KG |
|---|---|
| Study name / EAC code: | BIO MASTER.Cor Family / TA115 |
| Version and date of the Statistical Analysis Plan: | 3.0 from 18Mar2022 |
| Version and date of the underlying Clinical Investigation Plan: | Version 1-0 from 21Dec2018 |

| Print Name & Title | Signature | Date of Signature |
|--------------------------|-----------|-------------------|
| | | (DD MMM YYYY) |
| Clinical Project Manager | | |
| Scientist | | |
| Biostatistician | | |

# **Table of Content**

| Table of Con | tent | 2 |
|---|---|---|
| 0 Change | History | 2<br>5 |
| 1 Introduc | tion | 6 |
| 1.1 Aim | | 6 |
| 1.2 Dat | a for which quality control is required | 6 |
| 1.3 Ger | eral information | 6 |
| 2 Objectiv | es | 8 |
| 3 Investig | ational Device | 8 |
| 4 Study D | esign & Time Course | 9 |
| 5 General | Statistical Procedures | 11 |
| 5.1 Des | criptive analyses | 11 |
| 5.1.1 | Nominal – dichotomous data | 11 |
| 5.1.2 | Nominal data – more than two categories | 11 |
| | Scale / metric data | 12 |
| 5.1.4 | Ordinal data | 12 |
| 5.2 Infe | erential analyses | 13 |
| 5.3 Sigi | nificance level | 13 |
| 5.4 Miss | sing Data | 13 |
| | lusion of data from confirmatory data analysis | 13 |
| | groups | 14 |
| 5.7 Inte | erim analyses | 14 |
| 5.8 Soft | cware | 14 |
| 5.9 CDI | 1S export | 15 |
| 6 Specific | Study Dates | 16 |
| 6.1 Enr | ollment date | 16 |
| 6.2 Imp | plantation date | 16 |
| 6.3 Ter | mination date | 17 |
| 6.4 Cen | soring Date for Interim Analysis (not relevant for final analysis) | 18 |
| 7 Analysis | Sets | 19 |
| | Analysis Set | 19 |
| 7.2 Imp | plantation Analysis Set | 19 |
| 7.3 Cor | Family Analysis Set | 20 |
| 7.4 CR1 | Analysis Set | 21 |
| 7.5 CR1 | AutoAdapt Analysis Set | 21 |
| 7.6 AV | Opt Analysis Set | 22 |
| 7.7 Plex | a ProMRI S DX Analysis Set | 23 |
| 7.8 Inv | estigational Device Analysis Set | 23 |
| 7.9 Dat | a for a CONSORT diagram and CIR-chapter "study realization" | 24 |
| 7.9.1 | Number of patients | 24 |
| 7.9.2 | Study dates | 25 |
| 7.9.3 | Study duration | 25 |
| 7.9.4 | Premature termination | 26 |
| 7.9.5 | Investigational device not active | 27 |
| 8 General | data | 28 |
| 8.1 Ana | lysis set | 28 |
| 8.2 Var | iables | 28 |
| 8.2.1 | Baseline characteristics, medical history, and implantation | 28 |
| 8.2.2 | Assessment of ICD/CRT-D design (size and shape) | 37 |
| 8.2.3 | AV delay optimization feature (AV Opt) | 40 |
| 8.2.4 | Lead measurements (pacing thresh., sensing ampl., shock imp., lead imp.) | 42 |
| 8.2.5 | Sensing and pacing assessment | 45 |
| 8.2.6 | Arrhythmias and their treatment by the ICD/CRT-D system | 47 |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



reproduction or distribution is not permitted. Confidentiality:

This document and/or its contents are only for internal use.

| <b>BIO Master.Cor Family Version 3</b> | -0 |
|----------------------------------------|----|
| Cover Silect Statistical Alialysis F | IC |

| | 8.2.7 | Usage of Quick check | | 59 |
|---|---|---|---|---|
| | 8.2.8 | Assessment of statistic for ATP optimization | | 60 |
| | 8.2.9 | RV/LV active capture control at permanent DDI mode | | 60 |
| | 8.2.10 | MRI examinations, if performed independently from the study | | 61 |
| | 8.2.11 | Adverse Events (including assessment of causality – device or procedure relation | on) | 61 |
| | 8.2.12 | Device Deficiencies | | 61 |
| | 8.3 Trea | atment of Missing and Spurious Data | | 61 |
| | | usion of Particular Information | | 61 |
| | 8.5 Des | criptive Analyses | | 61 |
| | | otheses & Statistical Tests | | 61 |
| 9 | | | 62 | |
| | | lysis set | | 62 |
| | 9.2 Vari | ables | | 62 |
| | 9.2.1 | Handling assessment of Selectra catheter | | 62 |
| | 9.2.2 | Reports about cases with better CRT response using one of the new vectors | | 64 |
| | 9.2.3 | Usage and settings of MultiPole pacing (MPP) | | 65 |
| | 9.2.4 | Detailed information on SADEs related to MPP per event | | 67 |
| | 9.2.5 | Detailed information on SADEs related to the CRT AutoAdapt feature per event | | 68 |
| | 9.2.6 | Measurement of phrenic nerve stimulation, choice of tested vectors, finally | | |
| | | med settings and details on the use of the test page using LV VectorOpt | | 69 |
| | 9.2.7 | Programming of CRT AutoAdapt and overall assessment at 12-month follow-up | | 71 |
| | | atment of Missing and Spurious Data | | 72 |
| | | usion of Particular Information | | 72 |
| | | criptive Analyses | | 72 |
| | , , | otheses & Statistical Tests | | 72 |
| 1( | | | 73 | |
| | | lysis set | | 73 |
| | 10.2 Vari | | | 73 |
| | | Lead handling assessment | | 73 |
| | | Atrial sensing assessments | | 74 |
| | | Adverse events related to the Plexa S DX per event | | 75 |
| | 10.2.4 | , | | 76 |
| | | atment of Missing and Spurious Data | | 76 |
| | | usion of Particular Information | | 76 |
| | | criptive Analyses | | 76 |
| 4 . | | otheses & Statistical Tests ry Endpoint: Cor Family-related SADE-free rate until 3-month follow-up | 77 | 76 |
| Ι. | 11.1 Ana | · | // | 77 |
| | 11.1 Ana | • | | 78 |
| | | atment of Missing and Spurious Data | | 79 |
| | | usion of Particular Information | | 79 |
| | | criptive Analyses | | 79 |
| | | otheses & Statistical Tests | | 79 |
| 12 | | | 80 | |
| | | lysis set | - | 80 |
| | 12.2 Vari | | | 80 |
| | | atment of Missing and Spurious Data | | 81 |
| | | usion of Particular Information | | 81 |
| | | criptive Analyses | | 81 |
| | | otheses & Statistical Tests | | 81 |
| 13 | | | 82 | |
| | | lysis set | | 82 |
| | 13.2 Vari | | | 82 |
| | | atment of Missing and Spurious Data | | 84 |
| | | usion of Particular Information | | 84 |
| | 13.5 Des | criptive Analyses | | 84 |
| | 13.6 Hyp | otheses & Statistical Tests | | 84 |
| | | ning to this document are exclusively held | | , |
| by | BIOTRONIK | SE & Co. KG. Any non-authorized copying, | K | |

excellence for life

#### **Cover Sheet Statistical Analysis Plan** Page 4/88 **BIO|Master.Cor Family Version 3-0** Sec. Endpoint 3: CRT AutoAdapt feature (CRT only) 85 14.1 Analysis set 85 14.2 Variables 85 14.3 Treatment of Missing and Spurious Data 87 14.4 Exclusion of Particular Information 87 14.5 Descriptive Analyses 87 14.6 Hypotheses & Statistical Tests 87 Abbreviations 88 15



# **O Change History**

Version 1.0: Initial document.



# 1 Introduction

#### 1.1 Aim

The aim of this document is to provide detailed instructions on all mandatory descriptive and inferential statistical analyses for the Clinical Investigation Report (CIR).

#### 1.2 Data for which quality control is required

A quality control is needed for analyses of all endpoints(s) as defined in the clinical investigation plan (CIP) and referenced in this document.

#### 1.3 General information

The text contains verbatim excerpts from the CIP. Such excerpts are italicized with grey background; e.g.

. . . .

The main aspects and the design of the clinical investigation are presented in chapters 2 - 4

General statistical procedures are summarized in chapter 5. Those methods are used in case there is no other instruction within this document.

Definitions of the specific dates, e.g. effective randomization and termination are presented in chapter 6.

Specific analysis sets are defined in chapter 0.

Statistical analyses are handled in following chapters.

Thereby the following statistical considerations are specified:

- Definition of the analysis set for the following analyses, e.g. excluding patients without any measured or imputed data for this endpoint.
- Definition of the endpoint(s) to be analyzed including references to the source data, e.g. CRF sheet and item.
- Treatment of missing and spurious data for evaluation of the above endpoint(s).
- Exclusion of particular information from the evaluation of the above endpoint(s) in addition to the exclusion of patients from the analysis set.
- Descriptive analyses including tables and figures
- Statistical alternative hypothesis/hypotheses (HA) to analyze the above endpoint(s) if available.
- Statistical tests intended to analyze the above hypothesis/hypotheses if available.



All variables are defined in tables using the following columns:

Data file
 Name of a data file exported from the CDMS with one data row per unique identifier (e.g. patient specific "patient\_display\_ID\_full") additionally, a new data file ("SAR\_data") is generated by merging all relevant data from the original CDMS data files and generating derived variables (e.g. BMI from weight and height or date of first AE episode)

• Notes Information e.g. whether data has to be presented with descriptive

methods as defined in the following sub-chapter ("desc"),

as case listings or data needed for generating of derived variables only

("no report")

• Variable name Original name of a variable in the CDMS data file or

name of a derived variables (indicated with a suffix "\_SAR");

Variable label
 Original labels from the CDMS data will be used for generating the SAR

unless a new label is defined in this document ("NEW"); labels might be omitted or shortened ("...") if remaining clear

• Variable level Nominal, ordinal, scale (metric, continuous), text, or date

• Nominal values Original values from CDMS data will be used for generating the SAR

unless new nominal values are defined in this document ("NEW"); values might be omitted or shortened ("...") if remaining clear;

for numeric data this information is not applicable (n.a.)

| Data file, unique identifier patient_display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| patient_display_id_full | | | | | |
| Patient display ID | | | | | |
| nominal | | | | | |



# 2 Objectives

#### CIP chapter 7.1.Objectives

This study is designed as post market clinical follow-up study to identify and evaluate residual risks associated with the use of the Cor Family ICDs and the Plexa S DX lead that remained unrevealed even after risk analysis, risk mitigation and successful conformity assessment.

Moreover, the study aims at providing additional data, as required by regulatory authorities outside the CE-region. Furthermore, the performance and efficacy of the Cor Family devices and their features, as well as of the Plexa S DX lead shall be assessed. The results will be used for updating the clinical evaluation.

The primary objective of the clinical investigation is to confirm the clinical safety of the Cor Family ICDs by the analysis of the Cor Family-related SADEs until the 3-month follow-up.

Secondary objectives are the Kaplan-Meier estimate of the SADE-free rate at 3 and 12 months after implantation, the assessment of the automatic LV VectorOpt test, as well as the assessment of the CRT AutoAdapt feature.

# 3 Investigational Device

#### CIP chapter 4.1 Summary description of the device and its intended purpose

The investigational devices used in this clinical investigation are the ICDs and CRT-Ds of the Acticor/Rivacor ICD family and the Plexa ProMRI S DX ICD lead.

The ICDs/CRT-Ds of the Acticor/Rivacor family are state-of-the art implantable defibrillators intended for defibrillator therapy in patients with indication for primary or secondary prevention of sudden cardiac death. Triple-chamber devices (CRT-D) are additionally indicated for cardiac resynchronization therapy (CRT) for patients with congestive heart failure with ventricular asynchrony.

The Plexa ProMRI S DX ICD lead is intended for implantation in the right ventricle to deliver ATP and shock therapies during ventricular tachycardia. The lead provides sensing and pacing in the right ventricle, as well as sensing in the right atrium (floating atrial dipole).

Both the Acticor/Rivacor ICD family and the Plexa ProMRI S DX lead are equipped with a DF4 connector.

For better legibility in the following text, the investigational devices listed above are referred to as Cor Family ICDs and Plexa S DX lead, unless otherwise stated.



# 4 Study Design & Time Course

#### CIP chapter 8.1.4 Methods

During the course of the study, all clinical procedures are performed according to clinical routine. More detailed information can be found in the technical manual and in supporting study documents. The Automatic LV VectorOpt test for LV vector selection, and the AV Opt test or CRT AutoAdapt feature for AV delay optimization have to be used mandatorily in the respective devices unless contraindicated. The corresponding time schedule is described in section 9.1. All parameters and measurements that are recorded within the study are described in this section and are documented on the corresponding electronic Case listing forms (eCRFs). The investigator is required to use an electronic signature to approve the content of the data reported in the eCRFs. BIOTRONIK will monitor the content of the eCRFs as described in section 10. Data will be documented at the following points in time:

- -Enrollment/Baseline
- -Implantation
- -Pre-Hospital Discharge
- -3-month follow-up
- -6-month follow-up
- -12-month follow-up
- -Termination

The following events can be documented at any time:

- -Adverse Events
- -Device Deficiencies
- -Premature termination



#### CIP chapter 9.1 Overview

Table 5 : Overview of study procedures. The exact reference time for the 3-, 6- and 12-month follow-up is defined as 92 days, 183 days and 365 days after implantation, respectively. The applicable time window is  $\pm$  30 days around this reference time.

| Investigations | Enroll-<br>ment | Implan-<br>tation | PHD | 3-<br>Month<br>FU | 6-<br>Month<br>FU | 12-<br>Month<br>FU |
|---|---|---|---|---|---|---|
| Verification of in- and exclusion criteria | x | | | | | |
| Patient informed consent | x | | | | | |
| Documentation of<br>demographic and health<br>status data | x | | | | | |
| Documentation of<br>cardiovascular medication | х | х | x | × | × | x |
| Documentation of indication<br>for ICD/CRT-D therapy<br>(incl. available diagnostics) | X | | | | | |
| ICD/CRT-D implantation | | x | | | | |
| Assessment of ICD/CRT-D shape | | x | | | | |
| Assessment of Plexa S DX<br>Lead handling | | x | | | | |
| Assessment of Selectra<br>catheter handling | | x | | | | |
| Record device based<br>sensing, pacing threshold<br>and impedance values | | х | x | х | х | х |
| Evaluation of system<br>performance | | x | x | x | × | х |
| Evaluation of tachyarrythmia episodes | | x | X | x | x | x |
| Registration at HM Service<br>Center, hand out<br>CardioMessenger | | (x) | x | | | |
| Home Monitoring 'ON' | | x | x | x | x | (x) |
| Recording Episode IEGMs<br>(event triggered): 'ON' | | x | x | x | x | (x) |
| Automatic LV VectorOpt test | | (x) | x | (x) | | |
| CRT AutoAdapt 'ON'<br>(Acticor/Rivacor 7 CRT-D) | | (x) | x | (x) | (x) | (x) |
| Evaluation of CRT Auto<br>Adapt Feature (Acticor/<br>Rivacor 7 CRT-D) | | | | х | | (x) <sup>4</sup> |
| AV Opt Test (VR-T DX/<br>DR-T/Rivacor 5 CRT-D) | | | x | (x) | | |
| Documentation of Quick<br>Check | | | | x | x | X |
| Documentation of MPP<br>settings (for HF-T QP) | | x | x | × | × | × |
| Documentation of MRI examination | | | <u>x</u> | x | x | X |
| Assessment of patient's<br>wearing comfort (in case of<br>exchange) | | | | X | | |
| Evaluation of ATP statistics page | | | | | | x |
| eCRF completion | x | x | x | × | × | x |
| Provision of programmer data via ReportShare | | x | х | x | x | x |
| Adverse event and device deficiency reporting | x | X | x | × | x | X |
| Regular study termination | | | | | | x |

 $\underline{x}$ =if applicable, (x)=optional

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



# 5 General Statistical Procedures

# **5.1** Descriptive analyses

#### CIP chapter 11.1 Statistical design, method and analytical procedures

... For continuous variables descriptive statistics (mean, standard deviation, median, minimum, maximum and quartiles) will be calculated. For nominal variables absolute and relative frequencies will be calculated based on non-missing data. Ordinal variables are described similarly as continuous data (minimum, 1. quartile, median, 3. quartile, and maximum) or by absolute and relative frequencies based on non-missing data of each category.

For illustration, see the following standard tables with and without subgroup analyses based on dummy data.

#### 5.1.1 Nominal - dichotomous data

| Variable<br>(N total = 10) | | Category | N non-<br>missing | Absolute frequency | Relative<br>frequency<br>[%] |
|---|---|---|---|---|---|
| Sex | | Female | 9 | 5 | 55.6 |
| History of AF | | Yes | 8 | 4 | 50.0 |
| Variable<br>(N total = 10) | Category | Group<br>Randomization<br>group | N non-<br>missing | Absolute frequency | Relative<br>frequency<br>[%] |
| Sex | Female | Control<br>(N group = 3) | 3 | 2 | 66.7 |
| | | Therapy 1<br>(N group = 4) | 4 | 3 | 75.0 |
| | | All | 9 | 5 | 55.6 |
| History of AF | Yes | Control | 2 | 0 | 0.0 |
| | | Therapy 1 | 4 | 3 | 75.0 |
| | | All | 8 | 4 | 50.0 |

#### 5.1.2 Nominal data – more than two categories

| Variable (N total = 10) Patient self assessment at enrollment Patient self assessment at 12m FU | | N non-<br>missing | Very good<br>N(%) | Good<br>N(%) | Medium<br>N(%) | Poor<br>N(%) |
|---|---|---|---|---|---|---|
| | | 7 | 2 (28.6%) | 2 (28.6%) | 1 (14.3%) | 2 (28.6%) |
| | | 8 | 1 (12.5%) | 3 (37.5%) | 3 (37.5%) | 1 (12.5%) |
| Variable<br>(N total = 10) | Group<br>Randomization<br>group | N non-<br>missing | Very good<br>N(%) | Good<br>N(%) | Medium<br>N(%) | Poor<br>N(%) |
| Patient self assessment at enrollment | Control<br>(N group = 3) | 2 | 1 (50.0%) | 0 (0.0%) | 0 (0.0%) | 1 (50.0%) |
| | Therapy 1<br>(N group = 4) | 3 | 0 (0.0%) | 1 (33.3%) | 1 (33.3%) | 1 (33.3%) |
| | All | 7 | 2 (28.6%) | 2 (28.6%) | 1 (14.3%) | 2 (28.6%) |
| Patient self assessment at 12m FU | Control | 2 | 0 (0.0%) | 1 (50.0%) | 1 (50.0%) | 0 (0.0%) |
| | Therapy 1 | 4 | 0 (0.0%) | 2 (50.0%) | 1 (25.0%) | 1 (25.0%) |
| | All | 8 | 1 (12.5%) | 3 (37.5%) | 3 (37.5%) | 1 (12.5%) |



#### 5.1.3 Scale / metric data

| Variable<br>(N total = 10) | | N non-<br>missing | Mean | SD | Min | Lower quartile | Median | Upper<br>quartile | Max |
|---|---|---|---|---|---|---|---|---|---|
| Age [years] | | 7 | 51.7 | 15.0 | 25.0 | 40.0 | 57.0 | 60.0 | 70.0 |
| Height [cm] as measured at enro | llment | 8 | 177.3 | 14.4 | 150.0 | 170.0 | 179.0 | 187.5 | 195.0 |
| Variable<br>(N total = 10) | Group<br>Randomization<br>group | N non-<br>missing | Mean | SD | Min | Lower | Median | Upper<br>quartile | Max |
| Age [years] | Control<br>(N group = 3) | 2 | 55.0 | 7.1 | 50.0 | 50.0 | 55.0 | 60.0 | 60.0 |
| | Therapy 1<br>(N group = 4) | 3 | 56.7 | 15.3 | 40.0 | 40.0 | 60.0 | 70.0 | 70.0 |
| | All | 7 | 51.7 | 15.0 | 25.0 | 40.0 | 57.0 | 60.0 | 70.0 |
| Height [cm] as measured at enrollment | Control | 3 | 183.3 | 10.4 | 175.0 | 175.0 | 180.0 | 195.0 | 195.0 |
| | Therapy 1 | 3 | 175.0 | 21.8 | 150.0 | 150.0 | 185.0 | 190.0 | 190.0 |
| | All | 8 | 177.3 | 14.4 | 150.0 | 170.0 | 179.0 | 187.5 | 195.0 |

#### 5.1.4 Ordinal data

| Variable<br>(N total = 10) | N<br>missing | Min | Lower quartile | Median | Upper<br>quartile | Max |
|---|---|---|---|---|---|---|
| NYHA dass enrollment | 2 | 1.0 | 1.0 | 1.0 | 2.5 | 4.0 |
| NYHA dass 24m | 3 | 1.0 | 1.0 | 1.0 | 3.0 | 4.0 |

| Variable<br>(N total = 10) | Group<br>Randomization<br>group | N non-<br>missing | Min | Lower<br>quartile | Median | Upper<br>quartile | Max |
|---|---|---|---|---|---|---|---|
| NYHA dass enrollment | Control<br>(N group = 3) | 3 | 1.0 | 1.0 | 1.0 | 3.0 | 3.0 |
| | Therapy 1<br>(N group = 4) | 4 | 1.0 | 1.0 | 1.5 | 3.0 | 4.0 |
| | All | 8 | 1.0 | 1.0 | 1.0 | 2.5 | 4.0 |
| NYHA dass 24m | Control | 2 | 1.0 | 1.0 | 2.0 | 3.0 | 3.0 |
| | Therapy 1 | 3 | 1.0 | 1.0 | 2.0 | 4.0 | 4.0 |
| | All | 7 | 1.0 | 1.0 | 1.0 | 3.0 | 4.0 |



#### 5.2 Inferential analyses

#### CIP chapter 11.1 Statistical design, method and analytical procedures

To test the primary hypothesis an exact binomial tests is carried out. Additionally, an exact 2-sided 95% confidence interval will be generated.

#### 5.3 Significance level

#### CIP chapter 11.3 Level of significance and the power of the study

For the statistical test of the two-sided primary hypothesis, a two-sided p value less than 5% will be considered statistically significant.

No adjustment for multiple testing is foreseen, i.e. all analyses except those related to the primary end point were considered to be exploratory.

#### 5.4 Missing Data

#### CIP chapter 11.11 Handling of missing, unused and spurious data

Missing or spurious data will not be imputed.

Free text will be used to clarify other data.

Spurious data will be clarified via the query management, i.e. corrected after approval of an investigator. Remaining outliers will be identified during the review of the data before data base closure. In case of a clear evidence of a measurement error, the Statistical Analysis Plan will be updated in order to avoid any bias. Spurious data, which were not clarified by the query process before database closure, will be indicated. If appropriate, analyses will be performed both with /without such data.

#### 5.5 Exclusion of data from confirmatory data analysis

#### CIP chapter 11.12 Exclusion of data from the confirmatory data analysis

In the following cases, data are to be excluded from analysis or prevented from inclusion into analysis:

Exclusion of patients from the analysis set of the primary hypothesis:

- -No data is allowed to be collected and included in the absence of a documented informed consent.
- -Patients that are erroneously enrolled despite violation of inclusion or exclusion criteria at the time of enrollment
- -Patients without primary endpoint but premature study termination as defined for the primary endpoint are not included in the analysis set to avoid an over-estimation of the SADE-free rate.

Exclusion of data from patients included in the analysis set of the primary hypothesis:

- -Any event occurred later than the pre-specified time window after implantation as defined for the primary endpoint.
- -SADEs will be adjudicated by an internal adjudication board, whereby the seriousness and device relatedness will be re-examined. If any amply documented external physical influence (e.g. accident, sport, twiddling) or other causative AE led to the SADE, the SADE does not contribute to the endpoint.



#### 5.6 Subgroups

#### CIP chapter 11.9 Specification of subgroups

For this clinical investigation there is no specification of subgroups in the sense that analyses will be repeated for subsets of the pre-specified analysis set. However, there are different analysis sets defined for the primary and secondary endpoints.

#### 5.7 Interim analyses

#### CIP chapter 11.6 Level of significance and the power of the study

An interim analysis is planned after the completion of the 3-month follow-ups of all enrolled patients without prior study termination and final documentation of all prior primary endpoints. After this point in time, the data for testing the primary hypothesis will not be changed until the final analysis, and thus no multiplicity adjustment is required. Analysis of all other data and endpoints is explorative, therefore no multiplicity adjustment is required, either.

On request specific data might be provided to the competent authorities. Such kind of preliminary analysis would not bias the further data because no investigator except the Coordinating Investigator will be informed about the results. Except for safety reasons, no instruction for the further conductance of the clinical investigations will be made based on such preliminary analysis...

#### 5.8 Software

All analyses will be carried out using validated software, e.g. SAS version 9.4 or upgrades.



#### 5.9 CDMS export

The following data files are exported from the CDMS:

- event\_evaluation
- follow\_up\_3m
- follow\_up\_6m
- follow\_up\_12m
- adverse\_event
- auto\_lv\_vectoropt
- av\_opt
- baseline\_general
- cardiac diagnostic
- concomitant\_medication\_log
- deviation\_form\_bio
- deviation\_form\_bio\_log
- deviation\_form\_site
- device\_deficiency
- device\_log
- device\_log\_details
- enrollment
- hospitalization\_log
- implantation
- lead\_measurement
- medical\_history
- medication\_log\_details
- pre\_hospital\_dicharge
- tachyarrhythmia\_episode
- termination



# **6 Specific Study Dates**

#### 6.1 Enrollment date

#### CIP chapter 8.3.6. Point of enrolment and study termination

The point of enrollment is defined as the time of signature of the informed consent form by the patient. Study related procedures, documentation and collection/following of adverse events will start from this time on.

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| enrollment | DMICDT_i | Patient: Date of informed consent signature | date | n.a. |
| data_SAR | date_enrollment_SAR1 | Date of enrollment (PIC signature) | date | n.a. |

# 6.2 Implantation date

| Data file, identifier record_id & patient_display_id_full | | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|
| device_log_details | PRIMSTDT | Implantation/Use date | date | n.a. |

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| implantation | PRIMSTDT_i | Date of procedure (Implantation CRF) | date | n.a. |
| data_SAR | date_implantation_SAR <sup>2</sup> | Date of implantation | date | n.a. |





#### 6.3 Termination date

## CIP chapter 8.3.6 Point of enrolment and study termination

The point of study termination is defined as date of 12-month follow-up for patients with regular study termination.

The point of non-regular study termination can be the following:

- -Date of the last unsuccessful implantation attempt
- -Date of withdrawal of consent
- -Date of patient death
- -If patient is lost to follow-up, the date of last contact of the site study team (e.g. investigator or study nurse) with the patient
- -If patient is a drop-out for any other reason, the date of latest medical information of the patient (e.g. follow-up, IEGM)...

The above criteria are implemented as information for the investigator at the termination CRF. Thus, the date of study termination DSTRDT will be used until there is no contradiction to the date of a performed 12m follow-up.

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| follow_up_12m | $DSSUBNS \to$ | NEW 12mFU: Patient NOT SEEN for Follow-up | nominal | o True |
| | m12_DSSUBNS | | | o False |
| follow_up_12m | $SVFUSTDT_i \rightarrow$ | NEW 12mFU: Date of Follow-up | date | n.a. |
| | m12_SVFUSTDT_i | | | |
| termination | DSTRDT_i | Date of study termination | date | n.a. |
| data_SAR | date_termination_SAR3 | Minimum date of study termination or date of | date | n.a. |
| | | conducted 12m FU | | |



## 6.4 Censoring Date for Interim Analysis (not relevant for final analysis)

#### CIP chapter 8.1.4 Methods

Data will be documented at the following points in time:

- -Enrollment/Baseline
- -Implantation
- -Pre-Hospital Discharge
- -3-month follow-up
- -6-month follow-up
- -12-month follow-up
- -Termination

The following events can be documented at any time:

- -Adverse Events
- -Device Deficiencies
- -Premature termination

The censoring date is defined as the latest study procedure by which a previous AE should have been documented.

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| pre_hospital_discharge | $DSSUBNS \to$ | NEW PHD: Patient NOT SEEN for Follow-up | nominal | o True |
| | phd_DSSUBNS | | | o False |
| pre_hospital_discharge | $SVFUSTDT_i \rightarrow$ | NEW PHD: Date of Follow-up | date | n.a. |
| | phd_SVFUSTDT_i | | | |
| follow_up_3m | $DSSUBNS \to$ | NEW 3mFU: Patient NOT SEEN for Follow-up | nominal | o True |
| | m03_DSSUBNS | | | False |
| follow_up_3m | $SVFUSTDT_i \rightarrow$ | NEW 3mFU: Date of Follow-up | date | n.a. |
| | m03_SVFUSTDT_i | | | |
| follow_up_6m | $DSSUBNS \to$ | NEW 6mFU: Patient NOT SEEN for Follow-up | nominal | o True |
| | m06_DSSUBNS | | | ∘ False |
| follow_up_6m | $SVFUSTDT_i \rightarrow$ | NEW 6mFU: Date of Follow-up | date | n.a. |
| | m06_SVFUSTDT_i | | | |
| adverse_event | AESTDT_i | Onset date | date | n.a. |
| adverse_event | AEENDT_i | Date of resolution/Date of death | date | n.a. |
| device_deficiency | DERCDT_i | Date of detection | date | n.a. |
| data_SAR | date_implantation_SAR | Date of implantation or date of non-successful | date | n.a. |
| _ | | implantation attempt | | |
| data_SAR | date_termination_SAR | Date of conducted 12m FU or date of study | date | n.a. |
| | | termination | | |
| data_SAR | date_censoring_SAR4 | Date of censoring (latest date of AE onset, AE | date | n.a. |
| | | resolution, implantation, PHD, 3m FU, 6m FU, | | |
| | | 12m FU, or date of study termination) | | |







# 7 Analysis Sets

# 7.1 PIC Analysis Set

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| enrollment | DMICDT_i | Patient: Date of informed consent signature | date | n.a. |
| dat_SAR | analysis_set_signed_PIC_SAR <sup>5</sup> | Analysis set:PIC date available | nominal | ∘ Yes<br>∘ No |

## 7.2 Implantation Analysis Set

## CIP chapter 8.1.6 Replacement of subjects

During the course of the study, patients that drop out prior to any implantation attempt can be replaced as long as enrollment in the study is still ongoing. Patients who are not implanted with an investigational device and who did not come in contact with any investigational device during implantation attempt can also be replaced.

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| enrollment | DMICDT_i | Patient: Date of informed consent signature | date | n.a. |
| data_SAR | analysis_set_implantation_SAR6 | Analysis set Implantation (implantation or | nominal | o Yes |
| | | implantation attempt) | | ∘ No |





# 7.3 Cor Family Analysis Set

## CIP chapter 4.3 Model name including software version and accessories, table 1

Table 1: Eligible devices of the Cor Family

| Device name | Catalogue number |
|-------------------|------------------|
| Acticor 7 VR-T | |
| Acticor 7 VR-T DX | |
| Acticor 7 DR-T | |
| Acticor 7 HF-T | |
| Acticor 7 HF-T QP | |
| Rivacor 7 VR-T | |
| Rivacor 7 VR-T DX | |

| Data file, identifier record_id & patient_display_id_full | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|
| device_log_details | DIICDMDL | CRT-D model | nominal | o Acticor 7 HF-T o Acticor 7 HF-T QP o Rivacor 7 HF-T o Rivacor 7 HF-T QP o Rivacor 5 HF-T o Rivacor 5 HF-T o Rivacor 5 HF-T o Rivacor 5 HF-T QP |
| device_log_details | DIIDVMDL | ICD model | nominal | o Acticor 7 VR-T o Acticor 7 VR-T DX o Acticor 7 DR-T o Rivacor 7 VR-T o Rivacor 7 VR-T DX o Rivacor 7 DR-T o Rivacor 5 VR-T o Rivacor 5 VR-T o Rivacor 5 VR-T o Rivacor 5 DR-T o Rivacor 5 DR-T |

| | | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| enrollment | DMICDT_i | Patient: Date of informed consent | date | n.a. |
| | | signature | | |
| data_SAR | analysis_set_corfamily_SAR <sup>7</sup> | Analysis set Cor family: Acticor, | nominal | ∘ Yes |
| | | Rivacor implantation attempt | | o No |



# 7.4 CRT Analysis Set

| Data file, identifier record_id & patient_display_id_full | Variable<br>name | | Variable<br>level | Nominal values |
|---|---|---|---|---|
| device_log_details | DIICDMDL | CRT-D model | | o Acticor 7 HF-T o Acticor 7 HF-T QP o Rivacor 7 HF-T o Rivacor 7 HF-T QP o Rivacor 5 HF-T o Rivacor 5 HF-T o Rivacor 5 HF-T QP |

| signature date | n.a. |
|----------------|---------------|
| or HF nominal | ∘ Yes<br>∘ No |

## 7.5 CRT AutoAdapt Analysis Set

#### CIP chapter 8.1.4.9 CRT AutoAdapt (only Acticor 7 and Rivacor 7 CRT-Ds)

At implantation and/or Pre-Hospital Discharge CRT AutoAdapt shall mandatorily be programmed 'ON' in all CRT-D patients that are implanted with Acticor 7 or Rivacor 7, with the exception of patients with AV block, for whom this feature is contraindicated. (Note: CRT AutoAdapt is not available in Rivacor 5.)

| | | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|
| device_log_details | DIICDMDL | CRT-D model | | Acticor 7 HF-T Acticor 7 HF-T QP Rivacor 7 HF-T Rivacor 7 HF-T QP |

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| enrollment | DMICDT_i | Patient: Date of informed consent | date | n.a. |
| | | signature | | |
| data_SAR | analysis_set_CRTAutoAdapt_SAR9 | Analysis set AutoAdapt: Acticor 7 HF, | nominal | Yes |
| | | Rivacor 7 HF implantation attempt | | No |



## 7.6 AV Opt Analysis Set

<u>CIP chapter 8.1.4.5 AV delay optimization (for VR-T DX, DR-T, and Rivacor 5 HF-T and HF-T QP devices)</u>

For all patients with VR-T DX or DR-T devices (only if clinically indicated), and for patients with Rivacor 5 triple-chamber devices (as Rivacor 5 is not equipped with CRT AutoAdapt) with sinus rhythm of sufficient intrinsic rate, the AV Opt test has to be performed during the PHD follow-up. Performance of the test during the 3-month follow-up is acceptable if it was not done at PHD.

| Data file, identifier record_id & patient_display_id_full | Variable<br>name | | Variable<br>level | Nominal values |
|---|---|---|---|---|
| device_log_details | DIICDMDL | CRT-D model | nominal | o Rivacor 5 HF-T<br>o Rivacor 5 HF-T QP<br> |
| device_log_details | DIIDVMDL | ICD model | nominal | o Acticor 7 VR-T DX o Acticor 7 DR-T o Rivacor 7 VR-T DX o Rivacor 7 DR-T o Rivacor 5 VR-T DX o Rivacor 5 DR-T |

| Data file, identifier patient_display_id_full | | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|
| enrollment | DMICDT_i | Patient: Date of informed consent signature | date | n.a. |
| data_SAR | , | Analysis set AVopt: Rivacor 5 HF, Acticor DX,<br>Rivacor DX, Acticor DR, Rivacor DR<br>implantation attempt | | ∘ Yes<br>∘ No |



# 7.7 Plexa ProMRI S DX Analysis Set

#### CIP chapter 4.3 Model name including software version and accessories, table 2

Table 2: Eligible Plexa S DX leads

| Device name | Catalogue number |
|-------------------------|------------------|
| Plexa ProMRI S DX 65/15 | |
| Plexa ProMRI S DX 65/17 | |

| | | | Variable<br>level | Nominal values |
|---|---|---|---|---|
| device_log_<br>details | DIRVMDL | RV lead model | | o Plexa ProMRI S DX 65/15 o Plexa ProMRI S DX 65/17 |

| | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|
| enrollment | _ | Patient: Date of informed consent signature | date | n.a. |
| data_SAR | , = = = = | Analysis set Plexa: Plexa ProMRI S DX implantation attempt | | ∘ Yes<br>∘ No |

# 7.8 Investigational Device Analysis Set

| Data file, identifier patient_display_id_full | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|
| <u> </u> | , – – – | Analysis set investigational device: Acticor OR Rivacor OR Plexa ProMRI S DX implantation attempt | - | ∘ Yes<br>∘ No |

## 7.9 Data for a CONSORT diagram and CIR-chapter "study realization"

All analyses are performed for the PIC analysis set 13 if not mentioned otherwise.

#### 7.9.1 Number of patients

- Number of enrolled patients = number of patients in the PIC analysis set
- Number of enrollments per country from patient\_display\_id\_full
- Number of enrollments per investigational site from patient\_display\_id\_full
- Number of patients with implantation attempts = number of patients in the implantation analysis set
- Number of patients with implantation attempts of an investigational device= number of patients in the investigational device analysis set
- Number of patients with implantation attempts of a Cor family device= number of patients in the Cor Family analysis set
- Number of patients with implantation attempts of a Cor family CRT device= number of patients in the CRT analysis set
- Number of patients with implantation attempts of a Plexa ProMRI S DX lead = number of patients in the Plexa ProMRI S DX analysis set
- Number of patients with baseline<sup>14</sup>
- Number of patients with Pre-Hospital Discharge<sup>15</sup>
- Number of patients with 3mo FU<sup>16</sup>
- Number of patients with 6mo FU<sup>17</sup>
- Number of patients with 12mo FU<sup>18</sup>

| Data file, identifier patient display id full | | | | Nominal values |
|---|---|---|---|---|
| baseline_general | SVBLDT_i | Date of baseline assessment | date | n.a. |
| data_SAR | date_implantation_<br>SAR | Date of implantation | date | n.a. |
| pre_hospital_discharge<br>follow_up_3m<br>follow_up_6m<br>follow_up_12m | DSSUBNS → phd_DSSUBNS →m03_DSSUBNS →m06_DSSUBNS →m12_DSSUBNS | Patient NOT SEEN for Follow-up →Discharge Patient NOT SEEN for Follow-up → 03mFU: Patient NOT SEEN for Follow-up → 06m FU: Patient NOT SEEN for Follow-up → 12m FU: Patient NOT SEEN for Follow-up | nominal | o True<br>o False |
| pre_hospital_discharge<br>follow_up_3m<br>follow_up_6m<br>follow_up_12m | $\begin{array}{c} \text{SVFUSTDT} \\ \rightarrow \text{ phd\_SVFUSTDT} \\ \rightarrow \text{m03\_SVFUSTDT} \\ \rightarrow \text{m06\_SVFUSTDT} \\ \rightarrow \text{m12\_SVFUSTDT} \end{array}$ | Date of Follow-up →Discharge Date of Follow-up → 03mFU: Date of Follow-up → 06m FU: Date of Follow-up → 12m FU: Date of Follow-up | date | n.a. |





#### 7.9.2 Study dates

- Date of first-patient-in (FPI)
- Date of last-patient-in (LPI)
- Date of last-patient-out (LPO)

## 7.9.3 Study duration

Descriptive statistics to be reported for the PIC and for the implantation analysis set, respectively.

| Data file,<br>identifier<br>patient_<br>display id full | | | | | Nominal<br>values |
|---|---|---|---|---|---|
| data_SAR | descri<br>ptive | days_PIC_term_SAR <sup>19</sup> | Days from PIC to termination | scale | n.a. |
| _ | descri<br>ptive | days_implant_term_SAR <sup>20</sup> | Days from implantation attempt to termination | scale | n.a. |



#### 7.9.4 Premature termination

To be reported for the investigational PIC analysis set. 21

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | Notes | name | label | level | values |
| patient | | TIGITIC . | label | 10 4 01 | Tald Co |
| display_id_full | | | | | |
| 7 | | | | | |
| enrollment | case listings for | DMICDT | Patient: Date | data | n 2 |
| enrollment | case listings for<br>12m_SVFUSTDT = | DMICDI | of informed | uate | n.a. |
| | missing OR | | consent | | |
| | 12m_DSSUBNS = | | signature | | |
| data SAR | True | analysis_set_ | Analysis set | nominal | o Yes |
| uutu_0/t | | plexadx | of patients | | o No |
| | | _SAR | with Plexa | | |
| | | | ProMRI S DX | | |
| data CAD | - | | <br>Ali | | V |
| data_SAR | | analysis_set_<br>corfarm | of patients | | o Yes<br>o No |
| | | _SAR | with Acticor | | O NO |
| | | _5/1/ | or Rivacor | | |
| termination | 1 | DSTRDT | Date of study | date | n.a. |
| | | | termination | | |
| termination | | DSRTRM | Regular | nominal | |
| | | | study | | o No |
| termination | - | COETRREA | termination<br>Please | text | n 2 |
| termination | | COETRREA | specify | text | n.a. |
| | | | reason for | | |
| | | | early | | |
| | | | termination | | |
| termination | | DSETRREA | Reason for | nominal | o Patient moved away from investigational center |
| | | | early study | | o Patient is lost to follow-up |
| | | | termination | | o Patient withdrew consent to study participation |
| | | | | | o Patient death |
| | | | | | Judgement of physician Drop out according to protocol |
| | | | | | o Drop-out according to protocol<br>o Enrollment failure |
| | | | | | o Other |
| termination | Case listings for | DSSSDUSE | The patient | nominal | |
| | DSETRREA = | | allowed the | | o No / Not specified |
| | Patient withdrew | | further use | | |
| | consent to study | | of the | | |
| | participation | | already | | |
| | | | collected | | |
| | | | pseudonymiz<br>ed data | | |
| termination | Case listings for | DSDRPPRO | Please | nominal | o Patient is not implanted with a product of the |
| | DSETRREA = | | specify | | Cor Family of ICDs/CRT-Ds for any reason |
| | Drop-out | | "Drop-out | | o An explantation or replacement of the Cor |
| | according to | | according to | | Family ICD/CRT-D was performed |
| | protocol | | protocol" | | o Missing acceptance/compliance of the patient |
| | | | | | Significant worsening of general or pre-existing |
| | | | | | condition of the patient<br>o Other |
| termination | 1 | CODRPPRO | Please | text | n.a. |
| | | | specify | | |
| | | | "Drop-out | | |
| | | | according to | | |
| | | | protocol - | | |
| | ] | | Other" | | |



#### 7.9.5 Investigational device not active

| Data file, identifier | Notes | Variable | | Variable | Nominal values |
|---|---|---|---|---|---|
| patient_display_id_full | | name | label | level | |
| device_log_<br>details | Case listings for DTDVSTAT ≠Implante d and active | DTDVSTAT | Status of<br>device | nominal | <ul> <li>Implanted and active</li> <li>Deactivated but still connected and implanted</li> <li>Capped but still implanted</li> <li>Explanted and returned to manufacturer</li> <li>Explanted and discarded</li> <li>Attempted implantation, then returned to manufacturer</li> <li>Attempted implantation, then discarded</li> <li>Other</li> </ul> |
| | | PRIMSTDT | Implantation/<br>Use date | date | n.a. |
| | | DIICDMDL | CRT-D model | nominal | |
| | | DIIDVMDL | ICD model | nominal | |
| | | DIRVMDL | RV lead model | nominal | |



#### 8 General data

#### 8.1 Analysis set

The following analyses are performed for the investigational device analysis  $set^{22}$  and separately for the Plexa analysis  $set^{23}$ .

- Baseline characteristics and medical history
- Lead measurements
- Sensing and pacing assessment
- Adverse Events
- Device Deficiencies

The following analyses are performed for the Cor family analysis set<sup>24</sup>

- Assessment of ICD/CRT-D design
- Arrhythmias and their treatment by the ICD/CRT-D system
- Usage of QuickCheck
- Assessment of statistic for ATP optimization
- RV/LV active capture control at permanent DDI mode

The following analyses are performed for the AV Opt analysis set<sup>25</sup>

AV delay optimization feature

#### 8.2 Variables

#### 8.2.1 Baseline characteristics, medical history, and implantation

#### Baseline-general / Demographics

| Data file, identifier patient | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| display_id_full | | Harrie | label | ievei | values |
| baseline_general | descr. | DMSEX | Gender | nominal | ∘ Male |
| | | | | | o Female |
| | | | | scale | n.a. |
| data_SAR | descr. | DMAGE_65_SAR <sup>26</sup> | Age dichotomous greater | nominal | o Age >= 65 years |
| | | | than or equal 65 years | | o Age < 65 years |
| | descr. | DMAGE_75_SAR <sup>27</sup> | Age dichotomous greater | nominal | o Age >= 75 years |
| | | | than or equal 75 years | | o Age < 75 years |



#### Baseline-general / Physical examination

| Data file,<br>identifier patient_<br>display_id_full | | | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| baseline_general | descr. | VSHGHT | Height [cm] | scale | n.a. |
| | descr. | VSWGHT | Weight [kg] | scale | n.a. |
| | descr. | VSBMI | BMI [kg/m2] | scale | n.a. |
| | descr. | CVNYHA | Current NYHA classification | ordinal data | ∘ 1 |
| | | | | to be reported as nominal | ∘ 2 |
| | | | | variable | ∘ 3 |
| | | | | | ∘ 4 |

## Medical history / heart failure

| Data file,<br>identifier<br>patient_<br>display_id_<br>full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| medical_<br>history | descriptive | MHHF | History of heart failure | nominal | ∘ Yes ∘ No |
| | descriptive | MHHFE | Primary HF etiology | nominal | o Ischemic<br>o Non-ischemic |
| | descriptive | MHHFTYP | Type of HF | nominal | <ul><li>○ Left heart failure</li><li>○ Right heart failure</li><li>○ Global heart failure</li></ul> |
| | descriptive with "Unknown" to be analyzed as missing data | HOHF | Hospitalization for worsening of heart failure within the previous 12 months | nominal | ∘ Yes<br>∘ No<br>∘ Unknown |
| | No report | HOHFDT | Date of last hospitalization for heart failure | date | n.a. |
| | descriptive | days_hfhosp_<br>pic_SAR <sup>28</sup> | Days from last hospitalization for heart failure to PIC | scale | n.a. |
| | descriptive | MHCAD | History of coronary artery disease | nominal | ∘ Yes ∘ No |
| | descriptive for MHCAD = Yes | MHACCS | Prior acute coronary syndrome (any type) | nominal | ∘ Yes ∘ No |
| | descriptive | MHMI | Prior myocardial infarction | nominal | ∘ Yes ∘ No |
| | descriptive | PRRVC | Prior revascularization (PCI or CABG) | nominal | ∘ Yes ∘ No |



## Medical history / Brady- and tachyarrhythmias

| Data file, identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| medical_history | desciptive | MHSSS | History of sick sinus syndrome | nominal | ∘ Yes ∘ No |
| | descriptive | MHAVB | History of AV block | nominal | Yes ○ No |
| | descriptive for | MHAVBTYP | Type of AV block | nominal | o AV block I° |
| | MHAVB = Yes | | | | o AV block II° |
| | | | | | o AV block III° |
| | desciptive | MHBBB | History of bundle branch block | nominal | ∘ Yes / No |
| | desciptive for | MHBBBTYP | Type of bundle branch block | | o LBBB |
| | MHBBB = Yes | | | | o RBBB |
| | | | | | o Other |
| | desciptive | MHCNDDOT | History of other type of | nominal | ∘ Yes ∘ No |
| | | | conduction disease | | |
| | desciptive | MHAFB | History of atrial fibrillation | nominal | ∘ Yes ∘ No |
| | desciptive for | CVAFBTYP | Type of atrial fibrillation | nominal | o Paroxysmal |
| | MHAFB = Yes | | | | o Persistent |
| | | | | | <ul> <li>Long-standing persistent</li> </ul> |
| | | | | | o Permanent |
| | desciptive | MHAVA | History of other | nominal | ∘ Yes / No |
| | | | atria/supraventricular arrhythmias | | |
| | desciptive | MHVA | History of ventricular arrhythmia | nominal | ∘ Yes / No |

| Data file, identifier patient_display_id_full | | Variable<br>name | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| medical_history | l_history case listings<br>for MHBBBTYP = Other | | Specification of other type of bundle branch block | text | n.a. |
| | case listings<br>for MHCNDDOT = Yes | | Specification of other type of conduction disease | text | n.a. |
| | case listings<br>for MHAVA = Yes | | Specification of other atrial/supraventricular arrhythmias | text | n.a. |
| | case listings<br>for MHVA = Yes | COVA | Specification of history of ventricular arrhythmia | text | n.a. |



#### Medical history / Known comorbidities

| Data file, identifier patient_display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| medical_history | descriptive | MHCMB | Any Comorbidities known? | nominal | ∘ Yes ∘ No |
| | descriptive | MHHP | Hypertension (including well-controlled) | nominal | ○ Yes ○ No |
| | descriptive | MHVHD | Valvular heart disease | nominal | ∘ Yes ∘ No |
| | | MHAOVA | Aortic valve affected | nominal | ○ Yes ○ No |
| | Descriptive for | MHMIVA | Mitral valve affected | nominal | ∘ Yes ∘ No |
| | MHAOVA = Yes | MHMIIN | Mitral insufficiency | nominal | ∘ Yes ∘ No |
| | | MHMIST | Mitral stenosis | nominal | ◦ Yes ◦ No |
| | | MHTRVA | Tricuspid valve affected | nominal | ∘ Yes ∘ No |
| | | MHPUVA | Pulmonary valve affected | nominal | Yes ○ No |
| | descriptive | MHCVD | History of cerebrovascular disease (e.g. TIA / Stroke) | nominal | ∘ Yes ∘ No |
| | descriptive | MHPVAD | Peripheral vascular/arterial disease | nominal | ∘ Yes ∘ No |
| | descriptive | MHASTH | Asthma or other chronic lung disease (except COPD) | nominal | ∘ Yes ∘ No |
| | descriptive | MHCOPD | Chronic obstructive pulmonary disease (COPD) | nominal | ∘ Yes ∘ No |
| | descriptive | MHCKD | Chronic renal insufficiency / chronic kidney disease (CKD) (i.e. eGFR < 60) | nominal | ∘ Yes ∘ No |
| | descriptive | MHSAP | Sleep apnoea | nominal | ○ Yes ○ No |
| | descriptive for MHSAP = Yes | MHSAPTYP | Type of sleep apnoea | nominal | <ul><li>○ Central</li><li>○ Obstructive</li><li>○ Mixed</li></ul> |
| | descriptive | MHLIVR | Chronic liver disease | nominal | ∘ Yes ∘ No |
| | descriptive | MHDIAM | Diabetes mellitus | nominal | ∘ Yes ∘ No |
| | descriptive | MHANEM | Anemia | nominal | ∘ Yes ∘ No |
| | descriptive | MHCNCR | Cancer | nominal | ∘ Yes ∘ No |
| | descriptive | MHHPLP | Hyperlipidemia | nominal | ∘ Yes ∘ No |
| | descriptive | МНСМВОТН | Other comorbidities | nominal | ∘ Yes ∘ No |

| Data file, identifier patient_display id full | | | | | Nominal<br>values |
|---|---|---|---|---|---|
| | case listings | | Further specification of valvular heart disease (e.g. type, severity) | text | n.a. |
| | case listings<br>for MHCMBOTH<br>=Yes | СОСМВОТН | Specification of other comorbidities | text | n.a. |



# Cardiac diagnostic / ECG

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| cardiac_ | descriptive | EGHRT | Heart rate [bpm] | scale | n.a. |
| diagnostic | descriptive | CVEGARH | Atrial rhythm during ECG recording | nominal | <ul> <li>Sinus rhythm</li> <li>Atrial fibrillation</li> <li>Atrial flutter/other SVT</li> <li>Atrial paced rhythm</li> <li>Other</li> </ul> |
| | descriptive | CVEGVRH | Ventricular rhythm during ECG | nominal | o Intrinsic − atrial conduced<br>o Intrinsic − escape rhythm<br>o Ventricular paced rhythm<br>o Other |
| | descriptive for CVEGVRH ≠ ventricular paced rhythm | EGPRI | PR interval [ms] | scale | n.a. |
| | descriptive | EGQRS | QRS width (intrinsic) [ms] | scale | n.a. |
| | descriptive | EGQRSM | QRS morpholgy | nominal | o Normal o LBBB o RBBB o Indeterminate |

| Data file,<br>identifier<br>patient_<br>display id full | Notes | | | Nominal<br>values |
|---|---|---|---|---|
| cardiac_ | case listings<br>for CVEGARH = Other | Specification of other atrial rhythm during ECG recording | text | n.a. |
| | case listings<br>for CVEGVRH = Other | Specification of other ventricular rhythm during ECG recording | text | n.a. |

## Cardiac diagnostic / LVEF

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| cardiac_ | descr. | EHLVEF | Left ventricular ejection fraction [%] | scale | n.a. |
| diagnostic | | | | | |



#### Cardiac diagnostic / therapy indication

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| cardiac_<br>diagnostic | descr. | CECRT | CRT indication given | nominal | ∘ Yes<br>∘ No |
| | descr. | CECRTTYP | Type of CRT indication | nominal | CRT indication in sinus rhythm CRT indication in atrial fibrillation CRT indication and conventional pacing indication Other |
| | descr. | CEICDIND | ICD indication given | nominal | o Yes<br>o No |
| | descr. | CEICDTYP | Type of ICD indication | nominal | o Ventricular fibrillation (VF) o Symptomatic ventricular tachycardia (VT) o Asymptomatic ventricular tachycardia o Inducible VT/VF at EP study o Syncope o Primary prevention o Other |
| | descr. | CEBCINAS | Bradycardia indication given | nominal | o Yes<br>o No |
| | descr. | PRIM | Previous device implanted | nominal | o Yes<br>o No |
| | descr. | PRIMDVTY | Type pf previously implanted device | nominal | o Pacemaker o ICD o CRT pacemaker o CRT ICD o Implantable loop recorder |

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| cardiac_ | case listings | COEGVRH | Specification of other CRT indication | text | n.a. |
| diagnostic | for CECRTTYP = Other | | | | |
| | case listings | COICDOTH | Specification of other ICD indication | text | n.a. |
| | for CEICDTYP = Other | | | | |



#### **Baseline medication**

Medication is recorded on a continuous medication log documenting free text for trade names. An allocation between trade names and medication categories will be continuously maintained and updated at least during the blind review prior to any data analysis.

| Data file, identifier Notes | | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| record_id & | | name | label | level | values |
| patient_display_id_full | | | | | |
| medication_log_details | No report | CMBL | Baseline medication | nominal | Yes ○ No |
| | No report | CMTRT | Trade name | text | n.a. |

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| | descriptive | | BL med: ACE inhibitors | nominal | ∘ Yes ∘ No |
| | for CMBL = | aldost_block | BL med: Aldosterone blocker | nominal | ∘ Yes ∘ No |
| | Yes | angiotens_rec_block | BL med: Angiotensin receptor blocker | nominal | ∘ Yes ∘ No |
| | | antiarrhythmics | BL med: Antiarrhythmics | nominal | ∘ Yes ∘ No |
| | | anticoagulation | BL med: Anticoagulation | nominal | ∘ Yes ∘ No |
| | | antiplatelets | BL med: Antiplatelets | nominal | ∘ Yes ∘ No |
| | | betablocker | BL med: Betablocker (excluding sotalol) | nominal | ∘ Yes ∘ No |
| | | ccblocker | BL med: Calcium channel blocker | nominal | ○ Yes ○ No |
| | | digitalis | BL med: Digitalis | nominal | ○ Yes ○ No |
| | | diuretics | BL med: Diuretics (other than Aldosterone blocker) | nominal | ∘ Yes ∘ No |
| | | statins | BL med: Statins | nominal | ○ Yes ○ No |
| | | other_cv_med | BL med: Other cardiovascular medication | nominal | ∘ Yes ∘ No |
| | | non_cv_med | BL med: Non-cardiovascular medication | nominal | ∘ Yes ∘ No |



#### Implantation / investigational device system

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| implantation | descr. | PRIMTYP | Type of implantation | nominal | o De-novo system |
| | | | | | o Upgrade system |
| | | | | | o Device exchange |
| | descr. | PRIMRATY | Type of RA lead implantation | nominal | o New RA lead |
| | | | | | o Previously implanted RA lead |
| | | | | | o No RA lead implanted |
| | descr. | PRIMRVTY | Type of RV lead implantation | nominal | o New RV lead |
| | | | | | o Previously implanted RV lead |
| | | | | | o No RV lead implanted |
| | descr. | PRIMLVTY | Type of LV CS lead | nominal | o New LV CS lead |
| | | | implantation | | o Previously implanted LV lead |
| | | | | | ○ No attempt to implant LV CS lead |
| | | | | | <ul> <li>Unsuccessful attempt to implant LV CS lead</li> </ul> |
| | | | | | o No LV lead implanted |

| Data file,<br>identifier | Notes | Variable name | Variable<br>label | | Nominal values |
|---|---|---|---|---|---|
| patient_<br>display_id_full | | | | | |
| implantation | case listings<br>for PRIMLVTY = No<br>attempt to implant<br>LV CS lead | PRLVCSRE | Reason for no<br>attempt to<br>implant LV CS<br>lead | nominal | o Use of LV epicardial lead<br>o Use of LV endocardial lead<br>o Other |
| | | COLVCSRE | Specification of<br>other reason for<br>no attempt to<br>implant LV CS<br>lead | text | n.a. |
| | case listings<br>for PRIMLVTY =<br>Unsuccessful<br>attempt to implant<br>LV CS lead | PRIMLVRE | Main reason for<br>failure to implant<br>LV CS lead | | o Coronary sinus not identified o No suitable coronary vein identified o Extracardiac stimulation (e.g. n. phrenicus) o Other complication o LV lead deficiency o Other reason not related to a complication |
| | | COIMLVOT | Specification of other main reason for failure to implant LV CS lead | | n.a |
| | | PRIMLVP | Further attempts<br>to implant an LV<br>lead | nominal | <ul> <li>Endocardial LV lead planned/performed</li> <li>Epicardial LV lead planned/performed</li> <li>No LV lead planned</li> </ul> |

## Implantation/ Procedural data on LV CS lead implantation (only for CRT-D devices)

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| implantation | PRIMLVTY = New LV CS lead OR unsuccessful attempt to implant LV CS lead | PRLVVNG | Venogram performed prior to LV lead implantation | nominal | o Yes<br>o No<br>o Unknown |
| | | PRLVGCTH | Guide catheter used for LV lead implantation | nominal | o Yes<br>o No<br>o Unknown |
| | | PRLVGW | Guide wire used for LV lead implantation | nominal | o Yes<br>o No<br>o Unknown |
| | | PRLVSTL | Stylet used for LV lead implantation | nominal | o Yes<br>o No<br>o Unknown |


# Implantation / Usage of further accessories used

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| implantation | descriptive with "not applicable" OR "unknown" to be analyzed as missing data | | Used BIOTRONIK<br>accessories were | nominal | <ul> <li>Supplied with lead/device</li> <li>Obtained separately (NOT supplied with lead/device)</li> <li>Both Supplied with lead/device and Obtained separately</li> <li>Not applicable - no BIOTRONIK accessories have been used</li> <li>Unknown</li> </ul> |
| | descriptive for DUBACSUP = supplied obtained both case listings for DUBACPRB = Yes | COBACPRB | Did any problems with any used BIOTRONIK accessories occur Please specify the type of accessory and the | | <ul> <li>No - all used BIOTRONIK accessories were successfully used</li> <li>Yes - problems with used BIOTRONIK accessories have occurred</li> </ul> n.a. |
| | | | type of problem | | |

#### Implantation / Programmer type

| Data file, | Notes | | | Variable | |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| implantation | descriptive | DUPRGTYP | Programmer Type used | nominal | o Renamic |
| | | | | | o Renamic Neo |

# Implantation / initial devices (not restricted to investigational devices)

| Data file | Notes | | L. 1 - 1 - 7 - 7 | | Nominal<br>values |
|---|---|---|---|---|---|
| device_log_details | No report | PRIMSTDT | Implantation/Use date | date | n.a. |
| device_log_details | No report | DTEXDT | Explantation/deactivation date | date | n.a. |
| device_log_details | No report | DIDVTYP | General type of device | | o ICD<br>o CRT-D<br>o RA lead<br>o RV lead<br>o LV lead |
| device_log_details | Descriptive<br>for each<br>DIDVTYP | DIDVMDL | Device/lead model | text | n.a. |



#### 8.2.2 Assessment of ICD/CRT-D design (size and shape)

#### CIP chapter 8.1.4.5 Assessment of ICD/CRT-D design (size and shape)

The implanting investigator will be asked to assess the new design of the Cor Family devices ... In case of device exchanges, the patient will be asked about their wearing comfort compared to their previous device at the 3-month follow-up.

#### Implantation/ Assessment of ICD/CRT -D design

| Data file,<br>identifier<br>patient_display_<br>id_full | | | | | Ordinal<br>values |
|---|---|---|---|---|---|
| implantation | | DXIMLAS_R<br>DULDCAS | Required length of incision<br>Lead connection | nominal | o Very good<br>o Good |
| | descriptive | DULDBAS | Lead body leading out of the header | | o Adequate<br>o Poor<br>o Very poor |

| Data file,<br>identifier<br>patient_display_<br>id_full | | | | | Ordinal<br>values |
|---|---|---|---|---|---|
| implantation | case listings | COIMLAS | Please specify required length of incision | text | n.a. |
| | | COLDCAS | Please specify lead connection | text | n.a. |
| | | COLDBAS | Please specify lead body leading out of the header | text | n.a. |



#### Implantation/ Comparison of properties with BIOTRONIK's predecessor devices

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| implantation | descr. | DIPRDV | Provide information on predecessor devices | nominal | o Lumax o Idova o Iforia o Ilesto o Ilivia o Inlexa o Intica o Inventra o Iperia o Itrevia o Other |
| | descr. | DUPCMKAS | Ease / time needed for making the pocket for predecessor | nominal | <ul><li>Much more convenient</li><li>More convenient</li></ul> |
| | descr. | DUSZPHAS | Assessment of size and shape for the patient's comfort for predecessor | | o Similar<br>o Worse |
| | descr. | DUISPLAS01 | Ease, securing, and placement for predecessor | | ∘ Much worse |
| descr. DUCSI | | DUCSMTAS | Cosmetic outcome for predecessor | nominal | <ul><li>Much better</li><li>Better</li><li>Similar</li><li>Worse</li><li>Much worse</li></ul> |
| | descr. | DUPHSHAS | Interference for predecessor | nominal | <ul> <li>Much less (most physiological)</li> <li>Less (more physiological)</li> <li>Similar</li> <li>More (less physiological)</li> <li>Much more (least physiological)</li> </ul> |

| Data file, | Notes | Variable | Variable | Variable |
|---|---|---|---|---|
| identifier | | name | label | level |
| patient_ | | | | |
| display_id_full | | | | |
| | case listings<br>for DIPRDV =<br>Other | COPRDV | Please provide name of other predecessor device | text |
| | case listings | COPCMKAS | comment on ease/time needed for making the pocket for predecessor | text |
| | case listings | COSZPHAS | comment on assessment of size and shape for the patient' s comfort for predecessor | text |
| | case listings | COISPLAS01 | comment on ease, securing, and placement for predecessor | text |
| | case listings | COCSMTAS | comment on cosmetic outcome for predecessor | text |
| | case listings | COPHSHAS | comment on for predecessor | text |



#### Implantation/ Comparison of properties with competitor devices

| identifier patient_ | | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|
| ļ | | Provide information on most frequently used competitor device (Manufacturer) | | o Boston Scientific o Medtronic o Sorin Group / LivaNova o Abbott / St. Jude o Other o Unknown |
| | descriptive | Provide name of competitor device | nominal | |

| Data file,<br>identifier<br>patient_<br>display id full | | Variable<br>name | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| implantation | | DUPCMKAS01 | Ease / time needed for making the pocket for competitor | nominal | o Much more convenient<br>o More convenient |
| | descr. | USZPHAS01 | Assessment of size and shape for the patient's comfort for competitor | | o Similar<br>o Worse<br>o Much worse |
| | descr. | DUISPLAS02<br>NOTE deviating index | Ease, securing, and lead placement for competitor | | |
| | descr. | DUCSMTAS01 | Cosmetic outcome for competitor | nominal | <ul><li> Much better</li><li> Better</li><li> Similar</li><li> Worse</li><li> Much worse</li></ul> |
| | descr. | DUPHSHAS01 | Interference for competitor | nominal | <ul> <li>Much less (most physiological)</li> <li>Less (more physiological)</li> <li>Similar</li> <li>More (less physiological)</li> <li>Much more (least physiological)</li> </ul> |

| / | Notes | Variable | Variable | Variable |
|---|---|---|---|---|
| identifier | | name | label | level |
| patient_ | | | | |
| display_id_full | | | | |
| implantation | implantation case listings for DIDVMNF = Other | | Please provide name of "other" competitor | text |
| | case listings | | comment on ease/time needed for making the pocket for competitor | text |
| | case listings | COSZPHAS01 | comment on assessment of size and shape for the patient' s comfort for competitor | text |
| | J- | COISPLAS02 | comment on ease, securing, and placement for | text |
| | NOTE deviating index | | competitor | |
| | case listings | COCSMTAS01 | comment on cosmetic outcome for competitor | text |
| | case listings | COPHSHAS01 | comment on interference for competitor | text |

#### follow up 3m / Wearing Comfort in case of Device Exchange

| Data file,<br>identifier patient_<br>display_id_full | | | | Variable<br>level | Ordinal<br>values |
|---|---|---|---|---|---|
| implantation | no report | PRIMTYP | Type of implantation | | o De-novo system<br>o Upgrade system |
| follow_up_3m | descriptive for<br>PRIMTYP=Upgrade<br>system | | How did the patient assess the wearing comfort of the device compared to its predecessor | | <ul> <li>Much more convenient</li> <li>More convenient</li> <li>Similar</li> <li>Worse</li> <li>Much worse</li> </ul> |



#### 8.2.3 AV delay optimization feature (AV Opt)

<u>CIP chapter 8.1.4.5 AV delay optimization (for VR-T DX, DR-T, and Rivacor 5 HF-T and HF-T QP devices)</u>

For all patients with VR-T DX or DR-T devices (only if clinically indicated), and for patients with Rivacor 5 triple-chamber devices (as Rivacor 5 is not equipped with CRT AutoAdapt) with sinus rhythm of sufficient intrinsic rate, the AV Opt test has to be performed during the PHD follow-up. Performance of the test during the 3-month follow-up is acceptable if it was not done at PHD.

#### AV Opt test / AV delay optimization

| , | Notes | | | Variable | |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| av_opt | descriptive with | DUAVT | AV Opt test run | nominal | <ul> <li>Between Implantation and PHD</li> </ul> |
| | "Not done" to be | | | | o At PHD |
| | analyzed as | | | | o At 3-month Follow-up |
| | missing data | | | | o Not done |
| | descriptive | DUOAVT | Did the test suggest sensed | nominal | ∘ Yes |
| | | | and/or paced AV delay values? | | ∘ <b>No</b> |

| Data file, | Notes | Variable | Variable | Variabl | nominal |
|---|---|---|---|---|---|
| identifier | | name | label | е | values |
| patient_ | | | | level | |
| display_id_full | | | | | |
| av_opt | descriptive | DUAVTND01 | General lack of trust in automated test routines | nominal | <ul><li>o True ∘ False</li></ul> |
| | for DUAVT= | DUAVTND02 | Personal or institutional preference for use of alternative | nominal | <ul><li>o True ○ False</li></ul> |
| | Not done | DUAVTND03 | Patient conditions prescribe AV delay settings without | nominal | <ul><li>o True ○ False</li></ul> |
| | | | need for additional diagnostic aids | | |
| | | DUAVTND04 | Atrial fibrillation | nominal | <ul><li>o True ○ False</li></ul> |
| | | DUAVTND05 | No sufficient intrinsic rate | nominal | <ul><li>o True ○ False</li></ul> |
| | | DUAVTND10 | Other | nominal | <ul><li>o True ○ False</li></ul> |
| | | COAVTND | Please comment on reasons for not running AV Opt Test | text | n.a. |

| Data file,<br>identifier<br>patient_<br>display_id_full | | | | Variable<br>level | nominal<br>values |
|---|---|---|---|---|---|
| av_opt | descriptive | DUPCAVD | Suggested paced AV delay duration [ms] | scale | n.a. |
| | descriptive | DUSEAVD | Suggested sensed AV delay duration [ms] | scale | n.a. |



# AV Opt test / Final programmed AV delay settings

| Data file, | Notes | Variable | Variable | Variable | nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| av_opt | descr.* | DUAVDAP01 | AV Delay after pace 01 | scale | n.a. |
| | descr.* | DUAVDAP02 | AV Delay after pace 02 | scale | n.a. |
| | descr.* | DUAVDASE01 | AV Delay after sense 01 | scale | n.a. |
| | descr.* | DUAVDASE02 | AV Delay after sense 02 | scale | n.a. |
| | descr.* | DUHRT01 | AV Delay at rate 01 | scale | n.a. |
| | descr.* | DUHRT02 | AV Delay at rate 02 | scale | n.a. |
| | descr. | DUAVDCLA01 | NEW: Do you consider the <b>first</b> suggested AV delay clinically acceptable? | nominal | ∘ Yes ∘ No |
| | descr. | DUAVDCLA02 | NEW: Do you consider the <b>second</b> suggested AV delay clinically acceptable? | nominal | ∘ Yes ∘ No |
| | descr. | DUAVTOUT | NEW: Final programmed AV delay settings based upon the AV Opt test output | nominal | ∘ Yes ∘ No |
| | descr. | DUAVDPIP | Based upon the use of a personal/ institutional preference | nominal | ∘ Yes ∘ No |
| | descr. | DUAVDFUD | Based upon data from other follow-up affiliated diagnostics | nominal | ∘ Yes ∘ No |
| | descr. | DUAVDSPR | Adoption of values from the device's standard program | nominal | ∘ Yes ∘ No |
| | descr. | DUAVDIPR | Retention of AV delay settings from interrogated program | nominal | ∘ Yes ∘ No |
| | descr. | DUAVDVPC | Long AV delay to avoid ventricular pacing | nominal | ∘ Yes ∘ No |
| | descr. | DUAVDOTH | NEW: Other reason (please specify) for the final | nominal | ∘ Yes ∘ No |
| | | | programmed AV delay settings | | |

| Data file, | Notes | Variable | Variable | Variable | nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| av_opt | case listings for | COAVDREA01 | NEW: Reason for not considering <b>first</b> suggested | text | n.a. |
| | DUAVDCLA01 = No | | AV delay acceptable | | |
| | case listings for | COAVDREA02 | NEW: Reason for not considering <b>second</b> | text | n.a. |
| | DUAVDCLA02 = No | | suggested AV delay acceptable | | |
| | Case listing for | COAVDOTH | NEW: Please specify other reason for the final | text | n.a. |
| | DUAVDOTH = Yes | | programmed AV delay settings | | |

| Data file,<br>identifier<br>patient_<br>display id full | | Variable<br>name | | <br>Nominal<br>values |
|---|---|---|---|---|
| av_opt | descriptive | DUAVOTAS | How do you rate the AV Opt tool? | <ul><li>Very good</li><li>Good</li><li>Adequate</li><li>Poor</li><li>Very poor</li></ul> |

| Data file,<br>identifier<br>patient_<br>display_id_full | | | | Variable<br>level | nominal<br>values |
|---|---|---|---|---|---|
| _ ' | case listings for<br>DUAVOTAS = Poor OR<br>DUAVOTAS = Very poor | COAVOTAS | Please specify AV Opt tool rating | text | n.a. |





#### 8.2.4 Lead measurements (pacing thresh., sensing ampl., shock imp., lead imp.)

<u>CIP chapter 8.1.4.15 Lead measurements with Renamic programmer at implantation and each follow-up</u>

The system performance, i.e. appropriate sensing and pacing is evaluated at the end of the implantation procedure and at the end of each follow-up by either manually or automatically triggered lead measurements ...

The following "lead measurements" analyses have to be performed for implantation, Pre-Hospital Discharge, 3m follow-up, 6m follow-up, and 12m follow-up, whereby the variables labels have to

be indicated, respectively.

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| PRVISIT & | | | | | |
| patient_ | | | | | |
| display_id_full | | | | | |
| lead_ | No | PRVISIT | Visit | nominal | o Implantation |
| measurement | report | | | | <ul> <li>Pre-Hospital Discharge</li> </ul> |
| | | | | | o 3m Follow-up |
| | | | | | o 6m Follow-up |
| | | | | | o 12m Follow-up |

#### Lead measurements /Right Atrium (RA)

| | | | <del></del> | | |
|---|---|---|---|---|---|
| Data file | Notes | Variable | Variable | Variable | Nominal |
| PRVISIT & | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| lead_ | descr. | DURAMNA | No RA lead measurements available | nominal | o RA lead measurements not done |
| measurement | | | | | ○ RA lead not implanted/not active |
| | descr. | DURAMRH with | RA rhythm during sensing | nominal | o Sinus rhythm |
| | | "unknown" to be | measurements | | <ul><li>o Atrial fibrillation</li></ul> |
| | | analyzed as | | | <ul><li>o Atrial flutter/other SVT</li></ul> |
| | | missing data | | | <ul><li>o Atrial paced rhythm</li></ul> |
| | | and missing | | | o Other |
| | | data not | | | o Unknown |
| | | considered for | | | |
| | | percentages | | | |
| | descr. | DURASA | RA sensing amplitude [mV], mean | scale | n.a. |
| | | | value | | |
| | descr. | DURAPT | RA pacing threshold [V] | scale | n.a. |
| | descr. | DURAPTPW | Pulse width for RA pacing threshold | scale | n.a. |
| | | | measurements [ms] | | |
| | descr. | DURAPI | RA pacing impedance $[\Omega]$ | scale | n.a. |

#### Lead measurements / Right Ventricle (RV)

| Data file<br>PRVISIT &<br>patient_<br>display_id_full | Notes | | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| lead_<br>measurement | descr. | DURVMNA | No RV lead measurements available | nominal | <ul><li>○ RV lead measurements not done</li><li>○ RV lead not implanted/not active</li></ul> |
| | descr. | DURVMRH | RA rhythm during sensing measurements | nominal | <ul> <li>Intrinsic – atrial conducted</li> <li>Ventricular paced rhythm</li> <li>Other atrial conducted</li> <li>Ventricular paced rhythm</li> <li>Other</li> </ul> |
| | descr. | DURVSA | NEW: RV sensing amplitude [mV], mean value | scale | n.a. |
| | descr. | DURVPT | RV pacing threshold [V] | scale | n.a. |
| | descr. | | Pulse width for RV pacing threshold measurement [ms] | scale | n.a. |
| | descr. | DURVPI | RV pacing impedance $[\Omega]$ | scale | n.a. |
| | descr. | DURVSI | Painless shock impedance $[\Omega]$ | scale | n.a. |



#### Lead Measurements / Left Ventricle (LV)

| Data file<br>PRVISIT &<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| lead_<br>measurement | descr. | DULVMNA | No LV lead measurements available | nominal | o LV lead measurements not done<br>o LV lead not implanted/not active |
| | descr. | DULVTYP | type of LV lead | nominal | o Bipolar<br>o Quadripolar |
| | descr. | DULVSV | Permanently (first) programmed LV sensing vector | nominal | o LV1 tip to LV2 ring (bipolar) o LV1 tip to Can (unipolar) o LV2 ring to LV3 ring o LV2 ring to Can o LV3 ring to LV4 ring o LV3 ring to Can o LV4 ring to Can o LV4 ring to Can |
| | descr. | DULVPV01 | pacing vector | scale | o LV1 tip to LV2 ring o LV1 tip to LV3 ring o LV1 tip to LV4 ring o LV1 tip to RV coil/ring o LV1 tip to Can o LV2 ring to LV1 tip o LV2 ring to LV3 ring o LV2 ring to LV4 ring o LV2 ring to RV coil/ring o LV2 ring to Can o LV3 ring to LV1 tip o LV3 ring to LV1 tip o LV3 ring to LV1 tip o LV3 ring to LV1 tip o LV3 ring to LV4 ring o LV3 ring to LV4 ring o LV3 ring to RV coil/ring o LV3 ring to Can o LV4 ring to LV1 tip o LV4 ring to LV1 ring o LV4 ring to LV2 ring o LV4 ring to LV2 ring o LV4 ring to RV coil/ring o LV4 ring to RV coil/ring o LV4 ring to RV coil/ring o LV4 ring to RV coil/ring o LV4 ring to RV coil/ring |
| | descr. | DULVSA | (first) LV sensing amplitude [mV], mean value | scale | n.a. |
| | descr. | DULVPT01 | (first) LV pacing threshold [V] | scale | n.a. |
| | descr. | DULVPTPW01 | Pulse width for (first) LV pacing threshold measurements [ms] | scale | n.a. |
| | descr. | DULVPI01 | (first) LV pacing impedance $[\Omega]$ | scale | n.a. |

Lead measurements for the second vector are reported in chapter 9.2.3 Usage and settings of MultiPole pacing (MPP) .



| Data file patient_ display_id_full | | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|---|
| data_SAR | | type_SAR <sup>29</sup> | First pacing vector (New: LV1t-LV3r,<br>LV2r-LV3r, LV2r-C, LV3r-LV1t, LV3r-<br>C,LV4r-LV1t, LV4r-LV3r, LV4r-C) | | <ul><li>New vector</li><li>Old vector</li></ul> |
| _ | No report here- variable needed for MPP analysis | . <del></del> | Second pacing vector (New: LV1t-<br>LV3r,LV2r-LV3r,LV2r-C,LV3r-LV1t,<br>LV3r-C,LV4r-LV1t, LV4r-LV3r, LV4r-C) | - | <ul><li>New vector</li><li>Old vector</li></ul> |



All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



#### 8.2.5 Sensing and pacing assessment

# <u>CIP chapter 8.1.4.15 Lead measurements with Renamic programmer at implantation and each follow-up</u>

The investigator is asked to assess the sensing and pacing performance at the end of each follow-up...

#### Lead Measurements / System performance RA

| Data file<br>PRVISIT &<br>patient_<br>display_id_full | | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|---|
| lead_<br>measurement | descr. | DURASAAD | Adequate RA sensing | nominal | ∘ Yes ∘ No |
| | case listings for<br>DURASAAD = No | | Reason for inadequate RA sensing | | <ul><li>No intrinsic signal</li><li>Oversensing</li><li>Undersensing</li><li>Other</li></ul> |
| | descr. | DURAPCAD | Adequate RA pacing | nominal | ∘ Yes ∘ No |
| | case listings for DURAPCAD = No | | Reason for inadequate RA pacing | nominal | <ul> <li>No overpacing possible</li> <li>Exit block: no capture at maximum output</li> <li>Other</li> </ul> |

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| PRVISIT & | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| lead_ | case listings for | CORASAOT | Specification of other reason for inadequate RA | text | n.a. |
| measurement | DURASARE =Other | | sensing | | |
| | case listings for | CORAPCOT | Specification of other exit block for inadequate RA | text | n.a. |
| | DURAPCRE=Other | | pacing | | |

# Lead Measurements / System performance RV

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| PRVISIT & | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| lead_ | descr. | DURVSAAD | Adequate RV sensing | nominal | ∘ Yes ∘ No |
| measurement | descr. | DURASARE | Reason for inadequate | nominal | o No intrinsic signals |
| | | | RV sensing | | <ul><li>○ Oversensing</li></ul> |
| | | | | | <ul><li>o Undersensing</li></ul> |
| | | | | | o Other |
| | descr. | DURAPCAD | Adequate RV pacing | nominal | ∘ Yes ∘ No |
| | descr. | DURVPCRE | Reason for inadequate | nominal | ○ No overpacing possible |
| | | | RV pacing | | o Exit block: no capture at maximum output |
| | | | | | o Other |

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| PRVISIT & | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| lead_ | case listings for | CORVSAOT | Specification of other reason for inadequate RV | text | n.a. |
| measurement | DURVSARE=Other | | sensing | | |
| | case listings for | CORVPCOT | Specification of other exit block for inadequate RV | text | n.a. |
| | DURVPCRE=Other | | pacing | | |



# Lead Measurements / System performance LV

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| PRVISIT & | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| lead_ | descr. | DULVSAAD | Adequate LV sensing | nominal | ∨ Yes No |
| measurement | descr. | DULVSARE | Reason for inadequate | nominal | o No intrinsic signal |
| | | | LV sensing | | o Oversensing |
| | | | | | o Undersensing |
| | | | | | o Other |
| | descr. | DULVPCAD | Adequate LV pacing | nominal | ∘ Yes ∘ No |
| | descr. | DULVPCRE | Reason for inadequate | nominal | ○ No overpacing possible |
| | | | LV pacing | | <ul> <li>Exit block: no capture at maximum output</li> </ul> |
| | | | | | o Other |

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| PRVISIT & | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| lead_ | case listings for | COLVSAOT | Specification of other reason for inadequate LV | text | n.a. |
| measurement | DULVSARE=Other | | sensing | | |
| | case listings for | COLVPCOT | Specification of other exit block for inadequate LV | text | n.a. |
| | DULVPCRE=Other | | pacing | | |

#### 8.2.6 Arrhythmias and their treatment by the ICD/CRT-D system

#### CIP chapter 8.1.4.16 Tachyarrhythmia episodes

During the course of the study the following tachyarrhythmia episodes have to be recorded, analyzed and evaluated on the tachyarrhythmia episode form:

- All episodes detected in the VT-1, VT-2 or VF-zone
- All episodes with attempted and/or delivered therapies (ATP and/or shock)
- The first new and last two AF and/or SVT episodes between two follow-ups.

The appropriateness of the episode detection and the success of the delivered ATPs and/or shocks to terminate the episode will be evaluated...

#### **Detection zone and assessment**

| Data file<br>CEEPNUM | | Variable<br>name | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| tachy- | no report | CEEPNUM | Episode number | nominal | |
| | 5 x7 table CEEPLOC x<br>CEEPAS_corr_SAR | CEEPLOC | Detection zone | nominal | o nsVT/nsT o ATR o SVT o VT1 / VT2 o VF |
| | No report | CEEPAS | Episode<br>assessment | nominal | <ul> <li>○ AF</li> <li>○ Atrial flutter</li> <li>○ Sinus tachycardia</li> <li>○ Other SVT</li> <li>○ Non-sustained VT / VF</li> <li>○ Sustained VT / VF</li> <li>○ Oversensing / Other</li> </ul> |
| | 5 x7 table CEEPLOC x<br>CEEPAS_corr_SAR | CEEPAS_corr_SAR <sup>31</sup> | Episode<br>assessment -<br>corrected | nominal | o AF o Atrial flutter o Sinus tachycardia o Other SVT o Non-sustained VT / VF o Sustained VT / VF o Oversensing / Other |





#### Therapy in VF zone

| Data file<br>CEEPNUM | Notes | Variable<br>name | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| tachy-<br>arrhythmia_<br>episode | No report | DX1THAT01 | First therapy delivered | nominal | <ul><li>ATP one-shot</li><li>Shock</li><li>No therapy (shock charging aborted)</li></ul> |
| | | DXATPOSA01 | ATP one-shot successfully terminated the episode | nominal | o Yes<br>o No |
| | | DXSHKTOT01 | Number of shocks<br>delivered in VF zone | ordinal | n.a. |
| | | DXSHKAS01 | Shock(s) successfully terminated the episode in VF zone | nominal | o Yes<br>o No |
| | | CEEPOUT01 | Episode outcome in VF zone | nominal | <ul> <li>Spontaneously self-terminated</li> <li>Successful external defibrillation</li> <li>Patient death</li> <li>Other</li> </ul> |
| | | COEPOUT01 | Specification episode outcome in VF zone | text | n.a. |

# Therapy in VT zone

| - Inclupy III V | | | | | |
|---|---|---|---|---|---|
| Data file | Notes | Variable | Variable | | Nominal |
| CEEPNUM | | name | label | level | values |
| tachy-<br>arrhythmia_<br>episode | No report | DX1THAT02 | First therapy delivered in VT zone | nominal | o ATP o Shock o No therapy (shock charging aborted) |
| op.souc | | DXATPTOT02 | Number of ATP attempts in VT zone | nominal | . , |
| | | DXATPRES02 | ATP results in VT zone | nominal | <ul> <li>Episode terminated by ATP</li> <li>Shock(s) delivered after ATP failure</li> <li>No shock delivered after ATP failure</li> </ul> |
| | | DXSHKTOT02 | Number of shocks delivered in VT zone | ordinal | n.a. |
| | | DXSHKAS02 | Shock(s) successfully terminated the episode in VT zone | nominal | o Yes<br>o No |
| | | CEEPOUT02 | Episode outcome in <b>VT</b> zone | nominal | <ul> <li>Spontaneously self-terminated</li> <li>Successful external defibrillation</li> <li>Patient death</li> <li>Other</li> </ul> |
| | | COEPOUT02 | Specification episode outcome in <b>VT</b> zone | text | n.a. |



#### Appropriateness of episode detection per episode

Appropriateness of episode detection will be evaluated with respect to the consequences the detection has on the delivery of an ICD therapy.

- Detection zones that (may) result in delivery of a therapy (depending on the programming): VT1/VT2 or VF
- Detection zone that will never result in the delivery of a therapy: nsVT/nsT, ATR, or SVT
- Rhythm (episode assessment) that requires a therapy: sustained VT/VF and non-sustained
   VT/VF (with successful therapy; see below)
- Rhythm (episode assessment) that does not require a therapy: The remaining options for episode assessment and non-sustained VT/VF (without successful therapy, see below)

| | Rhythm that requires a therapy | Rhythm that does not require a therapy |
|---|---|---|
| ` ' ' ' ' | | Inappropriate detection (non-ventricular arrhythmia falsely detected; false positive) |
| result in the delivery of a therapy | | Appropriate detection (non-ventricular arrhythmia correctly detected; true negative) |



| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| tachy- | descriptive; | tp_episode_detection_SAR33 | Appropriate detection of ventricular | nominal | 0 1 |
| arrhythmia_ | case | | arrhythmia (true positive) | | o <b>0</b> |
| episode_SAR | listings for | fn_episode_detection_SAR34 | Inappropriate detection (ventricular | nominal | 0 1 |
| | all fn and fp | | arrhythmia not detected; false negative) | | o <b>0</b> |
| | episodes | tn_episode_detection_SAR35 | Appropriate detection (non-ventricular | nominal | 0 1 |
| | | | arrhythmia correctly detected; true negative) | | o <b>0</b> |
| | | fp_episode_detection_SAR36 | Inappropriate detection (non-ventricular | nominal | 0 1 |
| | | | arrhythmia falsely detected; false positive) | | o <b>0</b> |

The episode detection is evaluated by the following values:

- Sensitivity = sum tp / (sum tp + sum fn)
- Specificity = sum tn / (sum tn + sum fp)
- PPV = sum tp / (sum tp + sum fp)
- NPV = sum tn / (sum tn + sum fn)



All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



#### Appropriateness of episode detection per patient

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| _ | descri<br>ptive | ,_ , | Any tachy-arrhythmia episode with non-<br>missing information about the detection zone | nominal | ∘ Yes<br>∘ No |
| | | | Any tachy-arrhythmia episode with detection in the VT1/VT2 or VF zone | | ∘ Yes<br>∘ No |
| | | | All tachy-arrhythmia episodes with appropriate detection (all true positive or true negative) | nominal | ∘ Yes<br>∘ No |
| | | ,_ , | Any tachy-arrhythmia episode with inappropriate detection (any false positive or false negative) | nominal | ∘ Yes<br>∘ No |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



#### ATP efficacy per tp episode

Only applicable for true positive tachy-arrhythmia episodes<sup>41</sup> as defined before.

| | | | in a manufacture of the control of t | | |
|---|---|---|---|---|---|
| Data file | Notes | Variable | Variable | Variable | Nominal |
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| tachy- | descri | tpVF_ATP_SAR <sup>42</sup> | True positive episode in VF zone with ATP-one- | nominal | o <b>1</b> |
| arrhythmia_ | ptive | | shot therapy | | o <b>0</b> |
| episode_SAR | | tpVF_ATP_success_SAR43 | True positive episode in VF zone with successful | nominal | o <b>1</b> |
| | | | ATP-one-shot therapy | | o <b>0</b> |

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| tachy- | descri | tpVT_ATP_SAR <sup>44</sup> | True positive episode in VT1/VT2 zone with | nominal | ∘ 1 |
| arrhythmia_ | ptive | | at least one ATP therapy | | o <b>0</b> |
| episode_SAR | | tpVT_ATP_success_SAR <sup>45</sup> | True positive VT1/VT2 episode with | nominal | ∘ 1 |
| | | | successful ATP therapy | | o <b>0</b> |
| | | n_ATP_tpVT_SAR <sup>46</sup> | Number of ATP-attempts per true positive | Metric reported | ∘ 1 |
| | | | VT1/VT2 episode | as nominal | o <b>2</b> |

The ATP efficacy is evaluated by the following values:

- ATP VF efficacy rate = sum{VFtp\_ATP\_success\_SAR}/ sum{VFtp\_ATP\_SAR}
- ATP VT efficacy rate = sum{VTtp\_ATP\_success\_SAR}/ sum{VTtp\_ATP\_SAR}







#### ATP efficacy per patient (for tp episodes)

Only applicable patients with any true positive tachy-arrhythmia episodes<sup>47</sup> as defined before.

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| data_SAR | descri | any_tpVF_ATP_SAR <sup>48</sup> | Any true positive VF episode with ATP one- | nominal | o Yes |
| | ptive | | shot therapy | | o No |
| | | only_tpVF_noATP_SAR <sup>49</sup> | All true positive VF episodes without ATP | nominal | ∘ Yes |
| | | | one-shot therapy | | o No |
| | | only_tpVF_ATP_success_SAR <sup>50</sup> | All true positive VF episodes with ATP one- | nominal | ∘ Yes |
| | | | shot therapy were successful | | o No |
| | | any_tpVF_ATP_nosuccess_SAR <sup>51</sup> | Any true positive VF episode with delivered | nominal | o Yes |
| | | | but not successful ATP one-shot therapy | | o No |
| | | any_tpVT_ATP_SAR <sup>52</sup> | Any true positive VT episode with ATP | nominal | o Yes |
| | | | therapy | | o No |
| | | only_tpVT_noATP_SAR <sup>53</sup> | All true positive VT episodes without ATP | nominal | o Yes |
| | | | therapy | | o No |
| | | only_tpVT_ATP_success_SAR <sup>54</sup> | All true positive VT episodes with ATP | nominal | o Yes |
| | | | therapy were successful | | o No |
| | | any_tpVT_ATP_nosuccess_SAR <sup>55</sup> | Any true positive VT episode with delivered | nominal | ∘ Yes |
| | | | but not successful ATP therapy | | o No |

| • |
|-----------------------------------------|
| I |
| • |
| <u> </u> |
| l e e e e e e e e e e e e e e e e e e e |
| i |
| • |
| I |





#### Shock efficacy per tp episode

Only applicable for true positive tachy-arrhythmia episodes<sup>56</sup> as defined before.

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| tachy- | descri | tpVF_shock_SAR <sup>57</sup> | True positive episode in VF zone with at least | nominal | o <b>1</b> |
| arrhythmia_ | ptive | | one shock therapy | | ∘ 0 |
| episode_SAR | | tpVF_shock_success _SAR <sup>58</sup> | True positive episode in VF zone with | nominal | o <b>1</b> |
| | | | successful shock therapy | | ∘ 0 |
| | | n_shock_tpVF_SAR <sup>59</sup> | Number of shocks per true positive episode in | Metric | o <b>1</b> |
| | | | VF zone | reported | ∘ 2 |
| | | | | as nominal | |
| | | tpVT_shock_SAR <sup>60</sup> | True positive episode in VT zone with at least | nominal | o <b>1</b> |
| | | | one shock therapy | | o <b>0</b> |
| | | tpVT_shock_success _SAR <sup>61</sup> | True positive episode in VT zone with | nominal | o <b>1</b> |
| | | | successful shock therapy | | o <b>0</b> |
| | | n_shock_tpVT_SAR <sup>62</sup> | Number of shocks per true positive episode in | Metric | o <b>1</b> |
| | | | VT zone | reported | o <b>2</b> |
| | | | | as nominal | |

The shock efficacy is evaluated by the following values:

- Shock VF efficacy rate = sum{tpVF\_shock\_success\_SAR}/ sum{tpVF\_shock\_SAR}
- Shock VT efficacy rate = sum{tpVT\_shock\_success\_SAR}/ sum{tpVT\_shock\_SAR}



All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



# Shock efficacy per patient (for tp episodes)

Only applicable for patients with any true positive tachy-arrhythmia episodes<sup>63</sup> as defined before.

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| data_SAR | descri | any_tpVF_shock_SAR <sup>64</sup> | Any true positive VF episode with shock | nominal | o Yes |
| | ptive | | therapy | | o <b>No</b> |
| | | only_tpVF_noshock_SAR <sup>65</sup> | All true positive VF episodes without shock | nominal | ∘ Yes |
| | | | therapy | | o <b>No</b> |
| | | only_tpVF_shock_success_SAR <sup>66</sup> | All true positives VF episodes with shock | nominal | o Yes |
| | | | therapy were successful | | o No |
| | | any_tpVF_shock_nosuccess_SAR <sup>67</sup> | Any true positive VF episode with not | nominal | o Yes |
| | | | successful shock therapy | | o No |
| | | any_tpVF_shock_SAR <sup>68</sup> | Any true positive VT episode with shock | nominal | o Yes |
| | | | therapy | | o <b>No</b> |
| | | only_tpVF_noshock_SAR <sup>69</sup> | All true positive VT episodes without shock | nominal | o Yes |
| | | | therapy | | ∘ No |
| | | only_tpVF_shock_success_SAR <sup>70</sup> | All true positive VT episodes with shock | nominal | o Yes |
| | | | therapy were successful | | ∘ No |
| | | any_tpVF_shock_nosuccess_SAR <sup>71</sup> | Any true positive VT episode with not | nominal | o Yes |
| | | | successful shock therapy | | o No |

| <u> </u> |
|-------------|
| <del></del> |





# Therapy efficacy per patient (for tp episodes)

Only applicable for patients with any true positive tachy-arrhythmia episodes<sup>72</sup> as defined before.

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| data_SAR | descri | any_tpVF_therapy_SAR <sup>73</sup> | Any true positive VF episode with ATP or | nominal | o Yes |
| | ptive | | shock therapy | | o No |
| | | only_tpVF_therapy_success_SAR <sup>74</sup> | All true positive VF episodes with ATP or | nominal | o Yes |
| | | | shock therapy were successful | | o No |
| | | any_tpVF_therapy_nosuccess_SAR <sup>75</sup> | Any true positive VF episode with not | nominal | o Yes |
| | | | successful shock or ATP therapy | | o No |
| data_SAR | descri | any_tpVT_therapy_SAR <sup>76</sup> | Any true positive VT episode with ATP or | nominal | ∘ Yes |
| | ptive | | shock therapy | | ∘ No |
| | | only_tpVT_therapy_success_SAR <sup>77</sup> | All true positive VT episodes with ATP and | nominal | o Yes |
| | | | shock therapy were succesful | | ∘ No |
| | | any_tpVT_therapy_nosuccess_SAR <sup>78</sup> | Any true positive VT episode with not | nominal | o Yes |
| | | | successful ATP or shock therapy | | o No |



All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



### <u>Inappropriate therapies per fp episode</u>

Only applicable for false positive tachy-arrhythmia episodes<sup>79</sup> as defined before.

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| tachy- | descri | fp_episode_ATP_SAR80 | False positive episode with inappropriate | nominal | o <b>1</b> |
| arrhythmia_ | ptive | | ATP or ATP one-shot therapy | | o <b>0</b> |
| episode_SAR | | fp_episode_shock_SAR81 | False positive episode with inappropriate | nominal | o <b>1</b> |
| | | | shock therapy | | o <b>0</b> |
| | | fp_episode_ATP_shock_SAR82 | False positive episode with inappropriate | nominal | o <b>1</b> |
| | | | ATP, ATP-one-shot, or shock therapy | | ∘ 0 |

| Data file<br>patient_<br>display id full | | Variable<br>name | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| tachy-<br>arrhythmia_<br>episode_SAR | descri<br>ptive<br>or | | one-shot counts as 1) per false positive episode | as nominal | ○ 1<br>○ 2<br>○ |
| | listing | 11_3110ckp_cp130dc_3/1k | | as nominal | o 2<br>o |
| | | | | | ○ 1<br>○ 2<br> |







#### <u>Inappropriate therapies per patient (for fp episodes)</u>

Only applicable for patients with any false positive tachy-arrhythmia episodes<sup>86</sup> as defined before.

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| data_SAR | descri | any_fp_ATP_therapy_SAR <sup>87</sup> | Any false positive episode with inappropriate | nominal | o Yes |
| | ptive | | ATP therapy | | o No |
| | | any_fp_shock_therapy_SAR88 | Any false positive episode with inappropriate | nominal | o Yes |
| | | | ATP or shock therapy | | o No |
| | | any_fp_ATP_shock_therapy_SAR <sup>89</sup> | Any false positive VF episode with | nominal | o Yes |
| | | | inappropriate ATP or shock therapy | | o No |



All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



#### 8.2.7 Usage of Quick check

#### CIP chapter 8.1.4.11 Quick check

The use of QuickCheck is optional during the study...

The following analyses have to be performed for the 3m follow-up, 6m follow-up, and 12m follow-up, whereby the variables labels have to be indicated, respectively.

| Data file patient_ | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| display_id_full<br>follow_up_3m<br>follow_up_6m | descriptive | DUQCSUB | Was QuickCheck<br>used? | nominal | ∘ Yes ∘ No |
| follow_up_12m | descriptive<br>for DUQCSUB<br>= Yes | DUQCREA | Reason for<br>activation of<br>QuickCheck | nominal | <ul> <li>Routine check (instead of or in addition to scheduled HM follow-ups)</li> <li>Observation in Home Monitoring Data</li> <li>Home Monitoring Alert</li> <li>Patient demand (reassurance)</li> <li>Patient demand (symptoms)</li> <li>Other</li> </ul> |
| | | DUQCTRG | QuickCheck was<br>triggered | nominal | <ul> <li>While patient was on the phone</li> <li>After the patient has contacted the site</li> <li>After the site has contacted the patient</li> <li>Without patient contact</li> </ul> |
| | | DUQCTRGB | QuickCheck was<br>triggered by | nominal | <ul><li>Nurse</li><li>Physician</li><li>Cardiac technician</li><li>Other</li></ul> |
| | | _ | Was the QuickCheck transmission fast enough? | | o No<br>o No opinion |
| | descriptive | DUQCOAS | Overall assessment of the QuickCheck feature | nominal | o Very good o Good o Adequate o Poor o Very poor |

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| follow_up_3m | case listings for | COQCTRGB | Specification for Other Trigger for | text | n.a. |
| follow_up_6m | DUQCTRGB = Other | | QuickCheck | | |
| follow_up_12m | case listings | COQCOAS | Comment on Overall assessment of | text | n.a. |
| | for poor assessments | | QuickCheck | | |



#### 8.2.8 Assessment of statistic for ATP optimization

#### CIP chapter 8.1.4.17 Assessment of statistic for ATP optimization

If ATP optimization was programmed 'ON' (optional), the investigator will be asked to assess the statistics for ATP optimization at the 12-month follow-up for patients that experienced tachyarrhythmia episodes treated with ATP in the course of the study.

| Data file patient_ | Notes | | Variable<br>label | | Nominal values |
|---|---|---|---|---|---|
| display_id_full | | | | | |
| follow_up_12m | descriptive | DUATPON | Was ATP optimization programmed "on"? | nominal | ◦ Yes ◦ No |
| | descriptive for<br>DUATPON =Yes | | How was the comprehensibility of the new ATP Statistics page? | nominal | o Very good o Good o Adequate o Poor o Very poor |
| | Yes for<br>DUATPON =Yes | | How was the usefullness of the new ATP Statistics page? | nominal | <ul><li>Very good</li><li>Good</li><li>Adequate</li><li>Poor</li><li>Very poor</li></ul> |

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| follow_up_12m | case listings | COATPSAS01 | How was the comprehensibility of the new ATP | text | n.a. |
| | for poor | | Statistics page? | | |
| | assessments | COATPSAS02 | How was the usefullness of the new ATP Statistics | text | n.a. |
| | | | page? | | |

#### 8.2.9 RV/LV active capture control at permanent DDI mode

#### CIP chapter 8.1.4.18 RV/LV Capture Control at permanent DDI mode

Home Monitoring data will be analyzed to identify any patients in permanent DDI mode in whom capture control is activated in at least one of the ventricular channels (RV, LV and/or LV2). The AE database will be searched for Adverse Device Effects related to loss of capture that occurred in these patients.

Information for the CIR will be based on the Vigilance AE report and on separate Home Monitoring analyses.



#### 8.2.10 MRI examinations, if performed independently from the study

# CIP chapter 8.1.4.14 MRI examinations

If an MRI examination was performed during the course of the study (independently from the study), the following data will be recorded: Use of MRI AutoDetect, Use of MRI Test Mode, Adverse Events/Device Deficiencies related to the MRI procedure or activation of MRI AutoDetect.

The following case listings have to be reported for each 3m follow-up, 6m follow-up, or 12m follow-up with MRI scan performed since last follow-up.

Other information for the CIR will be based on the Vigilance AE report.

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| | no report | PRFUMRI | Routine MRI scan performed since last follow-up? | nominal | ∘ Yes ∘ No |
| follow_up_6m | case listings for | PRMRSTDT | Date of MRI scan | date | n.a. |
| follow_up_12m | PRFUMRI = Yes | | MRI AutoDetect feature used or attempted to be used | nominal | ∘ Yes ∘ No |
| | | PRMRADAS | MRI AutoDetect could be successfully programmed | nominal | ○ Yes ○ No |
| | | COMRADAS | Please specify | text | n.a. |
| | | | Was the 'MRI Test Mode' used to test the effect of programming the patient to MRI mode | nominal | ∘ Yes ∘ No |
| | | | Was deactivation of MRI mode checked via Home<br>Monitoring the day after the scan | nominal | ∘ Yes ∘ No |
| | | | Were any Adverse Events / Device Deficiencies detected in regard to the MRI AutoDetect? | nominal | ∘ Yes ∘ No |
| | | COSUM | General Comments | text | n.a. |

#### 8.2.11 Adverse Events (including assessment of causality – device or procedure relation)

Information for the CIR will be based on the Vigilance AE report.

#### 8.2.12 Device Deficiencies

Information for the CIR will be based on the Vigilance AE report.

#### 8.3 Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 8.4 Exclusion of Particular Information

See general definitions in chapter 5.5.

#### 8.5 Descriptive Analyses

See general definitions in chapter 5.1. and notes previous variable tables.

#### 8.6 Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 9 CRT Devices (HF-T and HF-T QP)

#### 9.1 Analysis set

All analyses are performed for the CRT analysis  $set^{90}$  or CRT AutoAdapt analysis  $set^{91}$  respectively.

#### 9.2 Variables

# 9.2.1 Handling assessment of Selectra catheter

# CIP chapter 8.1.4.14 Assessment of Selectra catheter handling (if applicable)

If a Selectra catheter (outer or outer and inner) is used to position the left ventricular lead, the implanting investigator will be asked to assess its features ...

#### Implantation / Usage of Selectra catheter and accessories

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| | descriptive | DUCTH | Was the Selectra catheter used? | nominal | o Yes<br>o No |
| | descriptive | | NEW: Please specify type(s) of <b>Selectra</b> catheter | - | <ul><li>Outer catheter</li><li>Outer and inner catheter</li></ul> |
| | descriptive for DUCTH=Yes | | NEW: Have there been any difficulties when using <b>specific Selectra</b> accessories? | nominal | o Yes<br>o No |
| | case listings for DUACCRAS01=Yes | | Please specify the difficulties when using Selectra accessories | text | n.a. |

| Data file,<br>identifier<br>patient_<br>display_id_full | | | | | Nominal<br>values |
|---|---|---|---|---|---|
| implantation | descriptive | DUSLTT | Slitter tool | nominal | ∘ True ∘ False |
| | for DUCTH=Yes | DUSRLL | Syringe with luer lock | nominal | ∘ True ∘ False |
| | | DUOWSC | One-way stop-cock | nominal | <ul><li>○ True ○ False</li></ul> |
| | | DUSGW | Seldinger guide wire | nominal | <ul><li>o True ∘ False</li></ul> |
| | | DUTRQR | Torquer | nominal | ∘ True ∘ False |
| | | DUSLCP | Sealing cap | nominal | ∘ True ∘ False |
| | | DUTVIT | Transval vularinsertion tool | nominal | <ul><li>o True ∘ False</li></ul> |
| | | DUBDCV | Bi -directional check valve | nominal | <ul><li>o True ∘ False</li></ul> |
| | | DUTBAD | Tuohy Borst Adapter (if available) | nominal | ∘ True ∘ False |



# Implantation / Assessment of Selectra and Selectra slitter tool handling

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|---|
| implantation | descriptive | DUTRQRAS | Torqueability | nominal | o Very good |
| | descriptive | DUFLXAS02 | Flexibility (distal end) | | o Good<br>o Adequate |
| | descriptive | DUGLDNAS | Gliding properties | | o Poor |
| | descriptive | DULDDLAS | Lead delivery | | ○ Very poor |
| | descriptive | DUSLTAAS | Slittability | | |
| | descriptive | DUXRVSAS03 | X-ray visibility | | |
| | descriptive | DUCTHAS | Overall handling of the catheter | | |
| | descriptive | DULDFXAS | Lead fixation mechanism | | |
| | descriptive | DUHNDSAS | Handling and design | | |
| | descriptive | DUSLTPAS | Slitting performance | | |
| | descriptive | DUSLTTAS | Overall handling of slitter tool | | |

| Data file,<br>identifier<br>patient_<br>display_id_full | | Variable<br>name | Variable<br>label | Variable<br>level | nominal<br>values |
|---|---|---|---|---|---|
| implantation | case listings | COTRQRAS | Please specify torqueability | text | n.a. |
| | for poor<br>assessments | COFLXAS02 | Please specify flexibility (distal end) | text | n.a. |
| | | COGLDNAS | Please specify gliding properties | text | n.a. |
| | | COLDDLAS | Please specify lead delivery | text | n.a. |
| | | COSLTAAS | Please specify slittability | text | n.a. |
| | | COXRVSAS03 | Please specify X-ray visibility | text | n.a. |
| | | COCTHAS | Please specify overall handling (catheter) | text | n.a. |
| | | COLDFXAS | Please specify lead fixation mechanism | text | n.a. |
| | | COHNDSAS | Please specify handling and design | text | n.a. |
| | | COSLTPAS | Please specify slitting performance | text | n.a. |
| | | COSLTTAS | Please specify overall handling (slitter tool) | text | n.a. |



#### Implantation / Usage of further accessories used

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| implantation | descriptive<br>with<br>"unknown" to<br>be analyzed as<br>missing data | | Used BIOTRONIK<br>accessories were | nominal | <ul> <li>Supplied with lead/device</li> <li>Obtained separately (NOT supplied with lead/device)</li> <li>Both Supplied with lead/device and Obtained separately</li> <li>Not applicable – no BIOTRONIK accessories have been used</li> <li>Unknown</li> </ul> |
| | DUBACSUP = o supplied o obtained o both | COBACPRB | Did any problems with any used BIOTRONIK accessories occur Please specify the type of accessory and the type of problem | | <ul> <li>No - all used BIOTRONIK accessories<br/>were successfully used</li> <li>Yes - problems with used BIOTRONIK<br/>accessories have occurred</li> </ul> n.a. |

#### Implantation / Programmer type

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| implantation | descriptive | DUPRGTYP | Programmer Type used | nominal | o Renamic |
| | | | | | o Renamic Neo |

#### 9.2.2 Reports about cases with better CRT response using one of the new vectors

#### CIP chapter 8.1.4.13 Improved CRT response after change of LV pacing vector

At the 6- and 12-month follow-up the investigator is asked to evaluate if a previous change of the LV pacing vector improved CRT response. The formerly used and the new vectors have to be documented.

The following analyses have to be performed for the 6m follow-up and 12m follow-up, whereby the variables labels have to be indicated, respectively.

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| follow_up_6m | descr. | DULVPVCH | Did you change the LV pacing vector(s) | nominal | ∘ Yes |
| follow_up_12m | | | during the last follow-up? | | o No |
| | descr. | CVCRTCHN | Did you observe a change in CRT response since last follow-up? | nominal | <ul><li>o Yes, improvement</li><li>o Yes, decrease</li><li>o No change</li></ul> |
| | descr. | CVLVVCRT | In your opinion, did the change of LV pacing vectors influence CRT response? | | <ul><li>Very likely</li><li>Likely</li><li>No opinion / not assessable</li><li>Unlikely</li><li>Very Unlikely</li></ul> |



#### 9.2.3 Usage and settings of MultiPole pacing (MPP)

#### CIP chapter 8.1.4.12 Usage and settings of MultiPole pacing (MPP)

The use of MultiPole Pacing (MPP) is optional within the study. However, if MPP was used in HF-T QP patients, the following data should be recorded: Programmed vectors, pacing thresholds, programmed pacing amplitudes, LV sensing polarity, sensing amplitude, LV-LV delay and LV-RV delay.

The following analyses have to be performed for the implantation, Pre-Hospital Discharge, 3m follow-up, 6m follow-up and 12m follow-up, whereby the variables labels have to be indicated, respectively.

#### <u>Lead measurements / Documentation of MPP settings</u>

| Data file,<br>identifier<br>PRVISIT &<br>patient_<br>display_id_full | Notes | | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| lead_<br>measurement | No report | PRVISIT | Visit | nominal | o Implantation<br>o Pre-Hospital Discharge<br>o 3m Follow-up<br>o 6m Follow-up<br>o 12m Follow-up |
| | descriptive | DUMPC | Was MultiPole Pacing used? | nominal | ∘ Yes ∘ No |
| | descriptive or case listings | DUPCORD | Pacing order | | o RV first<br>o LV first |
| | for | DULVLVD | LV-LV delay [ms] | scale | n.a. |
| | DUMPC=Yes | DUVVD | VV delay [ms] | scale | n.a. |
| | | DULVSA | (first) LV sensing amplitude [mV], mean value | scale | n.a. |

| Data file<br>PRVISIT &<br>patient_ | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| display_id_full | | | | | |
| lead_<br>measurement | descriptive or<br>case listings<br>for<br>DUMPC=Yes | DULVPT01 | Permanently programmed (first) LV pacing vector (first) LV pacing threshold [V] | | o LV1 tip to LV2 ring o LV1 tip to LV3 ring o LV1 tip to LV4 ring o LV1 tip to RV coil/ring o LV1 tip to Can o LV2 ring to LV1 tip o LV2 ring to LV3 ring o LV2 ring to LV4 ring o LV2 ring to RV coil/ring o LV2 ring to RV coil/ring o LV3 ring to LV1 tip o LV3 ring to LV1 tip o LV3 ring to LV1 ring o LV3 ring to LV2 ring o LV3 ring to LV2 ring o LV3 ring to LV4 ring o LV3 ring to RV coil/ring o LV3 ring to RV coil/ring o LV4 ring to LV1 tip o LV4 ring to LV1 tip o LV4 ring to LV2 ring o LV4 ring to LV2 ring o LV4 ring to RV coil/ring o LV4 ring to RV coil/ring o LV4 ring to RV coil/ring o LV4 ring to RV coil/ring o LV4 ring to RV coil/ring |
| | | DULVPTPW01 | Pulse width for (first) LV pacing | scale | n.a. |
| | | DULVPI01 | threshold measurements [ms] | scale | n.a. |
| data SAR | - | DULVPIO1 | (first) LV pacing impedance [Ω] First pacing vector (New: LV1t-LV3r, | | |
| data_JAK | | type_SAR | LV2r-LV3r, LV2r-C, LV3r-LV1t, LV3r-<br>C,LV4r-LV1t, LV4r-LV3r, LV4r-C) | nominal | o Old vector |



| D. L. Cl. | Int. L | M. 1.1.1. | M. 2.11. | V/- 1-1-1- | NI I |
|---|---|---|---|---|---|
| , | Notes | Variable | Variable | Variable | Nominal |
| identifier | | name | label | level | values |
| PRVISIT & | | | | | |
| patient_ | | | | | |
| display_id_full | | | | | |
| lead_ | | DULVPV02 | Programmed second LV pacing vector | nominal | o LV1 tip to LV2 ring |
| measurement | case listings | | | | o LV1 tip to LV3 ring |
| | for | | | | o LV1 tip to LV4 ring |
| | DUMPC=Yes | | | | o LV1 tip to RV coil |
| | | | | | o LV1 tip to ICD |
| | | | | | ○ LV2 ring to LV1 tip |
| | | | | | ○ LV2 ring to LV3 ring |
| | | | | | ○ LV2 ring to LV4 ring |
| | | | | | ○ LV2 ring to RV coil |
| | | | | | ○ LV2 ring to ICD |
| | | | | | o LV3 ring to LV1 tip |
| | | | | | ○ LV3 ring to LV2 ring |
| | | | | | o LV3 ring to LV4 ring |
| | | | | | ○ LV3 ring to RV coil |
| | | | | | o LV3 ring to ICD |
| | | | | | o LV4 ring to LV1 tip |
| | | | | | o LV4 ring to LV2 ring |
| | | | | | o LV4 ring to LV3 ring |
| | | | | | o LV4 ring to RV coil |
| | | | | | o LV4 ring to can |
| | | DULVPT02 | Second LV Pacing threshold [V] | scale | n.a. |
| | | DULVPTPW02 | Pulse width for second LV pacing | scale | n.a. |
| | | | threshold measurements [ms] | | |
| | | DULVPI02 | Second LV pacing impedance $[\Omega]$ | scale | n.a. |
| data_SAR | | DULVPV02 | Second pacing vector (New: LV1t- | nominal | o New vector |
| | | type SAR | LV3r,LV2r-LV3r,LV2r-C,LV3r-LV1t, | | ∘ Old vector |
| | | | LV3r-C,LV4r-LV1t, LV4r-LV3r, LV4r-C) | | |



#### 9.2.4 Detailed information on SADEs related to MPP per event

| Data file<br>identifier<br>record_id &<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| adverse_<br>event | case listings<br>for AEMPP =<br>Unlikely/Possible/P<br>robable/Causal<br>relationship AND | AEMPP | AE is related to MPP | nominal | o Not related o Unlikely o Possible o Probable o Causal relationship |
| | serious_ae_SAR =<br>Yes | serious_ae_ade_<br>SAR <sup>92</sup> | SA(D)E | nominal | ∘ Yes<br>∘ No |
| | | AEDVID | Please enter the related Device ID(s) from the Device Log below. Use "," to separate multiple entries. | nominal | |
| | | AESDTH | Event led to death | nominal | ∘ Yes<br>∘ No |
| | | AESLIFE | a life-threatening illness or injury | nominal | ○ Yes<br>○ No |
| | | AESDISAB | a permanent impairment of a body structure or body function | nominal | ∘ Yes<br>∘ No |
| | | AESHOSP | in-patient or prolonged hospitalization | nominal | ∘ Yes<br>∘ No |
| | | AESMIE | medical or surgical intervention<br>to prevent life-threatening<br>illness or injury or permanent<br>impairment to a body<br>structure/body function | nominal | ○ Yes<br>○ No |
| | | AESCONG | Event led to fetal distress, fetal death or a congenital abnormality or birth defect | nominal | ∘ Yes<br>∘ No |
| | | AEOUT | Outcome | nominal | <ul> <li>Resolved</li> <li>Resolved with</li> <li>sequelae</li> <li>Death</li> <li>Ongoing</li> <li>Ongoing at study</li> <li>termination</li> <li>Unknown</li> </ul> |
| | | COAEOUT | Please specify | text | n.a. |
| | | AEENDT_i | Date of resolution/Date of death | date | n.a. |
| data_SAR | Case listing as above | date_implantation<br>_SAR | Date of implantation | date | n.a. |





#### 9.2.5 Detailed information on SADEs related to the CRT AutoAdapt feature per event

| Data file identifier record_id & patient_ display_id_full | Notes | Variable<br>name | Variable<br>label | level | Nominal<br>values |
|---|---|---|---|---|---|
| adverse_<br>event | Note misspelling "possbile" case listings | AECRTAUA | AE is related to CRT AutoAdapt | nominal | o Not related o Unlikely o Possbile o Probable o Causal relationship |
| | for AECRTAUA = Unlikely/Possible/ | serious_ae_SAR | SA(D)E | nominal | ∘ Yes<br>∘ No |
| | Probable/Causal relationship AND serious_ae_SAR | AEDVID | Please enter the related Device ID(s) from the Device Log below. Use "," to separate multiple entries. | nominal | |
| | = Yes | AESDTH | Event led to death | nominal | <ul><li>Yes</li><li>No</li></ul> |
| | | AESLIFE | a life-threatening illness or injury | nominal | <ul><li>Yes</li><li>No</li></ul> |
| | | AESDISAB | a permanent impairment of a body structure or body function | nominal | ∘ Yes<br>∘ No |
| | | AESHOSP | in-patient or prolonged<br>hospitalization | nominal | ∘ Yes<br>∘ No |
| | | AESMIE | medical or surgical intervention to<br>prevent life-threatening illness or<br>injury or permanent impairment to a<br>body structure/body function | nominal | ∘ Yes<br>∘ No |
| | | AESCONG | Event led to fetal distress, fetal death or a congenital abnormality or birth defect | nominal | ∘ Yes<br>∘ No |
| | | AEOUT | Outcome | nominal | <ul> <li>Resolved</li> <li>Resolved with</li> <li>sequelae</li> <li>Death</li> <li>Ongoing</li> <li>Ongoing at study</li> <li>termination</li> <li>Unknown</li> </ul> |
| | | COAEOUT | Please specify | text | n.a. |
| data_SAR | | AEENDT_i<br>date_implantation<br>SAR | Date of resolution/Date of death Date of implantation | date<br>date | n.a.<br>n.a. |



9.2.6 Measurement of phrenic nerve stimulation, choice of tested vectors, finally programmed settings and details on the use of the test page using LV VectorOpt

#### Chapter 7.2.2.2 Secondary endpoint 2: Automatic LV VectorOpt test (CRT only)

... Furthermore, the choice of tested vectors, the number of performed PNS threshold measurements, the finally programmed settings and details on the use of the test page will be recorded as further data of interest ...

#### Automatic LV VectorOpt Test

| Data file identifier patient_display_id_full | | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|
| auto_lv_<br>vectoropt | descriptive | Automatic LV VectorOpt test done at | nominal | o PHD<br>o Implantation<br>o 3-month Follow-Up |
| | descriptive | Did you perform the RV-LV conduction time test? | nominal | <ul><li>Yes, only RVp-LVs</li><li>Yes, only RVs-LVs</li><li>Yes, both: RVp-LVs and RVs-LVs</li><li>No</li></ul> |
| | case listings<br>for<br>COLVVTND<br>not missing | Please specify not performing<br>Auto LVVectorOpt test | text | n.a. |

# Automatic LV VectorOpt Test / Manual and automatic testing of pacing vectors

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| auto_lv_ | descriptive | DUNVST | Number of vectors selected | ordinal | |
| vectoropt | | | for testing (minimum 3) | | |
| | descriptive | DUBOTHM | Were both measurements performed with | nominal | ∘ Yes |
| | | | the same subset of vectors? | | ∘ No |
| | case listings | СОВОТНМ | Please specify difference of tested vectors | text | n.a. |
| | for DUBOTHM | | | | |
| | = No | | | | |



#### Automatic LV VectorOpt Test / Manual and automatic testing of pacing vectors / HF-T QP

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| auto_lv_ | descr. | DULVVTF01 with "not | Was the automatic LV | nominal | ∘ Yes |
| vectoropt | | done" to be analyzed | VectorOpt test performed | | ○ No, other number tested |
| | | as missing data | for all 20 vectors | | o Not done |
| | descr. | DUNVST01 | NEW: Other number of | ordinal | |
| | | | vectors tested <>20 | | |
| | descr. | DULVTHAT01 | Time needed to run Auto | scale | n.a. |
| | | | LV threshold measurement | hh:mm:ss has to be | |
| | | | for 20 or selected vectors | converted to min | |

# Automatic LV VectorOpt Test / Manual and automatic testing of pacing vectors / HF-T

| Data file identifier patient_display_id_full | | | | | Nominal<br>values |
|---|---|---|---|---|---|
| auto_lv_<br>vectoropt | | done" to be analyzed | Was the automatic LV<br>VectorOpt test performed<br>for all 5 vectors | | <ul><li>o Yes</li><li>o No, other number tested</li><li>o Not done</li></ul> |
| | descr. | | NEW: Other number of vectors tested <b>&lt;&gt;5</b> | ordinal | |
| | descr. | | LV threshold measurement | scale<br>hh:mm:ss has to be<br>converted to min | n.a. |

# Automatic LV VectorOpt Test / PNS measurement

| Data file identifier patient_display_id_full | | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|---|
| auto_lv_ | descr. | DUPNSNVS | Number of vectors for which the PNS threshold was measured | ordinal | |
| vectoropt | descr. | DUPNSPPV | PNS threshold of finally programmed pacing vector [V] | scale | n.a. |

#### Automatic LV VectorOpt Test / Assessment

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| auto_lv_ | descriptive with "Not | DURVLVA | Do you consider | nominal | ∘ Yes |
| vectoropt | done" to be analyzed | S | the RV-LV | | o No |
| | as missing data | | conduction time | | o Not done |
| | | | test helpful? | | |
| | descriptive | DUPRSPV | Preselection of | nominal | ○ Selection of vector in programmer table |
| | | | the pacing | | Selection of 'Setting' button |
| | | | vectors for the | | o Using toggle buttons |
| | | | test was done by | | <ul> <li>Choosing from the LV pacing polarity window</li> </ul> |
| | | | | | o Other means |

| Data file,<br>identifier<br>patient_<br>display_id_full | | | | Variable<br>level | nominal<br>values |
|---|---|---|---|---|---|
| auto_lv_ | case listings for | COPRSPV | Please specify other means | text | n.a. |
| vectoropt | DUPRSPV =Other means | | for preselection of pacing vectors | | |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



#### 9.2.7 Programming of CRT AutoAdapt and overall assessment at 12-month follow-up

#### CIP chapter 8.1.4.9 CRT AutoAdapt (only Acticor 7 and Rivacor 7 CRT-Ds)

At implantation and/or Pre-Hospital Discharge CRT AutoAdapt shall mandatorily be programmed 'ON' in all CRT-D patients that are implanted with Acticor 7 or Rivacor 7, with the exception of patients with AV block, for whom this feature is contraindicated. (Note: CRT AutoAdapt is not available in Rivacor 5.)

#### <u>CIP chapter 7.2.2.3 Secondary endpoint 3: CRT AutoAdapt (CRT only)</u>

... Furthermore, information on the programming of the feature and an overall assessment at the 12-month follow-up (if applicable) contribute to the further data of interest ...

The following analyses have to be performed for the 12m follow-up data. 93 94

| Data file,<br>identifier<br>PRVISIT &<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| measurement | no<br>report | PRVISIT | Visit | nominal | o 12m Follow-up |
| | descr. | DUAUAON | NEW: CRT AutoAdapt "ON" at the end of the 12mFU | nominal | ∘ Yes ∘ No |
| | descr. | DUADAVRD | Adaptive AV reduction | nominal to<br>be reported<br>as ordinal<br>data | ○ 0.5<br>○ 0.6<br>○ 0.7<br>○ 0.8<br>○ 0.9 |
| | descr. | DUADAVLL | Adaptive AV lower limits [ms] | | o50 o60 o70 o80 o90<br>o100m o110m o120m<br>o130m o140m o150m |
| | descr. | DUVPC | Ventricular pacing | nominal | o BiV<br>o RV<br>o LV |
| | descr. | DUICPH | Initially paced chamber | nominal | ∘ RV<br>∘ LV |
| | descr. | DUVVDAVP | VV delay afer Vpace [ms] | scale | n.a. |
| | descr.* | DUAVDAP | AV Delay after pace 01 | scale | n.a. |
| | descr.* | DUAVDAP01 | AV Delay after pace 02 | scale | n.a. |
| | descr.* | DUAVDASE | AV Delay after sense 01 | scale | n.a. |
| | descr.* | DUAVDASE01 | AV Delay after sense 02 | scale | n.a. |
| | descr. | DUMCRTP | Mean CRT pacing since last follow-up [%] | scale | n.a. |
| | descr. | DUAVDAPO | Optimized AV delay after pace [ms] | scale | n.a. |
| | descr. | DUAVDASO | Optimized AV delay after sense [ms] | scale | n.a. |

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| PRVISIT & | | | | | |
| patient_ | | | | | |
| display_id_full | | | | | |
| lead_ | descr. | COAUAON for | Please specify why CRT AutoAdapt "OFF" or "AV Adapt" | text | n.a |
| measurement | | DUAUAON = No | | | |


The following analyses have to be performed for the 12m follow-up data. 95 96

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| follow_up_12m | no report | DUAUAON | CRT AutoAdapt "ON" | nominal | ∘ Yes |
| | | | | | ○ No |
| | descriptive | DUPRGAS | Programmability | nominal | ∘ Very easy |
| | for DUAUAON | | | | ∘ Easy |
| | = Yes | | | | o Adequate |
| | | | | | o Difficult |
| | | | | | ○ Very difficult |
| | | | Clinical acceptability | nominal | ∘ Very good |
| | | | of the algorithm's decision | | ∘ Good |
| | | | | | o Adequate |
| | | | | | o Poor |
| | | | | | o Very poor |
| | | DUAUAOAS | Overall assessment of the | nominal | o Very good |
| | | | CRT AutoAdapt feature | | ∘ Good |
| | | | | | o Adequate |
| | | | | | o Poor |
| | | | | | o Very poor |

| Data file<br>patient_<br>display_id_full | | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|---|
| | case listings | COPRGAS | Comment on programmability | text | n.a. |
| | for poor assessments | | comment on clinical acceptability of the algorithm's decision | text | n.a. |
| | | COAUAOAS | comment on overall assessment | text | n.a. |

#### 9.3 Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

See Automatic LV VectorOpt Test / Manual and automatic testing of pacing vectors / HF-T QP.

See <u>Automatic LV VectorOpt Test / Assessment.</u>

#### 9.4 Exclusion of Particular Information

See general definitions in chapter 5.5.

#### 9.5 Descriptive Analyses

See general definitions in chapter 5.1 and notes previous variable tables.

#### 9.6 Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



#### 10 Plexa ProMRI S DX

#### 10.1 Analysis set

All analyses are performed for the Plexa ProMRI S DX analysis set<sup>97</sup>

#### 10.2 Variables

#### 10.2.1 Lead handling assessment

CIP chapter 8.1.4.6 Assessment of Plexa S DX lead handling (if applicable)

During implantation, the handling of the Plexa S DX lead will be assessed by the implanting physician.

#### Implantation / Assessment of Plexa Pro MRI S DX lead handling

| Data file, identifier patient_display_id_full | | Variable<br>name | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| implantation | descr. | DUFLXAS01 | Flexibility of the Plexa ProMRI S DX | nominal | o Very good<br>o Good<br>o Adequate |
| | descr. | DUPSHAS | Push-ability of the Plexa ProMRI S DX | | o Poor |
| | descr. | DUPSBHAS | Positioning behavior of the Plexa ProMRI S DX | | <ul><li>Very poor</li></ul> |
| | descr. | DUERBHAS | Extension/retraction behavior of the Plexa ProMRI S DX screw | | |
| | descr. | DUXRVSAS01 | X-ray visibility of the extended screw of the Plexa ProMRI S DX | | |
| | descr. | DUFXBHAS | Fixation behavior of the Plexa ProMRI S DX | | |
| | descr. | DUXRVSAS02 | X-ray visibility of the Plexa ProMRI S DX in its final position | | |
| | descr. | DUSTLHAS | Stylet handling in regard to the Plexa ProMRI S DX? | | |

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | nominal<br>values |
|---|---|---|---|---|---|
| implantation | case<br>listings | COFLXAS01 | Please specify flexibility of the Plexa ProMRI S DX | text | n.a. |
| | case<br>listings | | Please specify the push-ability of the<br>Plexa ProMRI S DX | text | n.a. |
| | case<br>listings | | Please specify the positioning behavior of the Plexa ProMRI S DX | text | n.a. |
| | case<br>listings | | Please specify extension/retraction behavior of the Plexa ProMRI S DX screw | text | n.a. |
| | case<br>listings | | Please specify X-ray visibility of the extended screw of the Plexa ProMRI S DX | text | n.a. |
| | case<br>listings | | Please specify fixation behavior of the<br>Plexa ProMRI S DX | text | n.a. |
| | case<br>listings | | Please specify X-ray visibility of the<br>Plexa ProMRI S DX in its final position | text | n.a. |
| | case<br>listings | | Please specify stylet handling in regard to the Plexa ProMRI S DX | text | n.a. |



#### 10.2.2 Atrial sensing assessments

#### Lead Measurements / System performance RA

The following analyses have to be performed for implantation, pre-hospital\_ discharge, 3m follow-up, 6m follow-up, and 12m follow-up, whereby the variables labels have to be indicated,

respectively.

| respectively. | | | | | |
|---|---|---|---|---|---|
| Data file,<br>identifier<br>PRVISIT &<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
| lead_<br>measurement | no report | PRVISIT | Visit | nominal | o Implantation o Pre-Hospital Discharge o 3m Follow-up o 6m Follow-up o 12m Follow-up |
| | descriptive | DURASAAD | Adequate RA sensing | nominal | ∘ Yes<br>∘ No |
| | descriptive | DURASARE | Reason for inadequate RA sensing | nominal | <ul><li>No intrinsic signal</li><li>Oversensing</li><li>Undersensing</li><li>Other</li></ul> |



#### 10.2.3 Adverse events related to the Plexa S DX per event

| Data file | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| record id & | | | | | |
| patient_ | | | | | |
| display_id_full | | | | | |
| data_SAR | case listings for | imp_PRIMSTDT | Date of procedure (Implantation | date | n.a. |
| data_5/110 | the data below | | CRF) | uutc | ii.u. |
| device_log_ | No report | DIRVMDL | RV lead model | nominal | |
| details | но тероге | record id | Record ID | nominal | |
| | No report | | Please enter the related Device | | ••• |
| adverse_ | мо герогі | AEDVID | | nominal | |
| event | | | ID(s) from the Device Log below. | | |
| | | | Use "," to separate multiple | | |
| | | | entries. | | |
| | case listings for | AERELIDV | AE is related to the | nominal | ∘ Not related |
| | AEDVID = | | investigational device | | o Unlikely |
| | record_id with | | | | o Possible |
| | DIRVMDL | | | | o Probable |
| | contains "Plexa" | | | | <ul> <li>Causal relationship</li> </ul> |
| | and DIRVMDL | AERELIPR | AE is related to the | nominal | ○ Not related |
| | contains "DX" | | investigational device procedure | | o Unlikely |
| | | | | | o Possible |
| | NOTE that | | | | o Probable |
| | AEDVID may | | | | <ul> <li>Causal relationship</li> </ul> |
| | contain multiple | AESLIFE | a life-threatening illness or injury | nominal | ∘ Yes |
| | device IDs | | | | ∘ No |
| | | AESDISAB | a permanent impairment of a | nominal | ∘ Yes |
| | | | body structure or body function | | ∘ No |
| | | AESHOSP | in-patient or prolonged | nominal | ∘ Yes |
| | | | hospitalization | | ∘ No |
| | | AESMIE | medical or surgical intervention | nominal | ∘ Yes |
| | | | to prevent life-threatening illness | | ∘ No |
| | | | or injury or permanent | | - |
| | | | impairment to a body | | |
| | | | structure/body function | | |
| | | AESCONG | Event led to fetal distress, fetal | nominal | ∘ Yes |
| | | , | death or a congenital abnormality | | ∘ No |
| | | | or birth defect | | |
| | | AEOUT | Outcome | nominal | ∘ Resolved |
| | | | | oiiiidi | <ul> <li>Resolved with sequelae</li> </ul> |
| | | | | | o Death |
| | | | | | o Ongoing |
| | | | | | o Ongoing at study |
| | | | | | termination |
| | | | | | o Unknown |
| | | COAEOUT | Please specify | text | n.a. |
| | | AEENDT | Date of resolution/Date of death | date | n.a. |
| | | ALLINDI | pate of resolution/pate of death | uale | II.a. |



#### 10.2.4 Early detection of atrial fibrillation (episodes)

| Data file identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| record_id & | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| tachyarrhythmia_ | descriptive | CVAFON | New onset of AF | nominal | ∘ Yes |
| episode | | | | | ∘ No |
| | descriptive | CEFUAFHM | AF episode detected | nominal | ∘ Yes |
| | | | by Home Monitoring | | ∘ No |
| | and 2x2 table | | prior to follow-up visit | | |
| | CVAFON x CEFUAFHM | | | | |

#### 10.3 Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 10.4 Exclusion of Particular Information

See general definitions in chapter 5.5.

#### 10.5 Descriptive Analyses

See general definitions in chapter 5.1 and notes previous variable tables.

#### 10.6 Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 11 Primary Endpoint: Cor Family-related SADE-free rate until 3-month follow-up

#### 11.1 Analysis set

All analyses are performed for the Cor family analysis set<sup>98</sup> excluding the following patients:

#### CIP chapter11.12 Exclusion of data from confirmatory data analysis

Exclusion of patients from the analysis set of the primary hypothesis:

- -No data is allowed to be collected and included in the absence of a documented informed consent<sup>99</sup>
- -Patients that are erroneously enrolled despite violation of inclusion or exclusion criteria at the time of enrollment<sup>100</sup>
- -Patients without primary endpoint but premature study termination as defined for the primary endpoint  $^{101}$

## <u>CIP chapter</u> 7.2.1 <u>Primary endpoint and hypotheses: Cor Family-related SADE-free rate until 3-month follow-up</u>

The following patients are not included in the analysis set for this endpoint:

Patients without endpoint but premature study termination before or exactly at 61 days after implantation (3 months defined as 92 days after implantation – 30 days would still be in accordance to the CIP) are not included in the analysis set to avoid an over-estimation of the SADE-free rate.



#### 11.2 Variables

<u>CIP chapter</u> 7.2.1 <u>Primary endpoint and hypotheses: Cor Family-related SADE-free rate until 3-month follow-up</u>

SADEs will be adjudicated by an internal adjudication board, whereby the seriousness and device relatedness will be re-examined. If any amply documented external physical influence (e.g. accident, sport, twiddling) or medical AE caused the SADE, it does not contribute to this endpoint.

| Data file<br>record_id &<br>patient_<br>display_id_full | | | | | Nominal<br>values |
|---|---|---|---|---|---|
| event_<br>evaluation | no report | AESTDT | Onset date | date | n.a. |
| event_<br>evaluation | no report | AERELSET <sup>102</sup> | Adverse Event is relevant for SADE endpoint | nominal | <ul><li>Yes</li><li>No</li></ul> |
| event_<br>evaluation | no report | AERELPET <sup>103</sup> | Adverse Event is relevant for primary endpoint | nominal | <ul><li>Yes</li><li>No</li></ul> |

| record_id & patient_ | Notes | | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| display_id_full | | | | | |
| data_SAR | no report | date_implantation_SAR | Date of implantation | date | n.a. |
| data_SAR | no report | | Date of censoring (latest date of AE onset, AE resolution, implantation, PHD, 3m FU, 6m FU, 12m FU, or date of study termination) | date | n.a. |
| data_SAR | descriptive & inferential | | Any primary endpoint within the prespecified time-period | nominal | <ul><li>Yes</li><li>No</li></ul> |





See general definitions in chapter 5.4.

#### 11.4 Exclusion of Particular Information

<u>CIP chapter 7.2.1 Primary endpoint and hypotheses: Cor Family-related SADE-free rate until 3-month follow-up</u>

SADEs will be adjudicated by an internal adjudication board, whereby the seriousness and device relatedness will be re-examined. If any amply documented external physical influence (e.g. accident, sport, twiddling) or medical AE caused the SADE, it does not contribute to this endpoint. SADEs that occur later than the 3-month follow-up, and SADEs with onset date later than or exactly at 123 days after implantation (3 months defined as 92 days after implantation + 30 days would still be in accordance to the CIP) in case the 3-month follow-up was not conducted or conducted outside the specified time interval do not contribute to this endpoint.

#### 11.5 Descriptive Analyses

See general definitions in chapter 5.1 and notes previous variable tables.

#### 11.6 Hypotheses & Statistical Tests

<u>CIP chapter 7.2.1 Primary endpoint and hypotheses: Cor Family-related SADE-free rate until 3-month follow-up</u>

The safety of the Cor Family ICDs will be evaluated by asking the investigator to record any adverse event. While all adverse events have to be recorded throughout the study, only the Serious Adverse Device Effects (SADE) possibly or securely related to the Cor Family devices (SADE- $d_{Cor}$ ) until 3-month follow-up are counted for this primary endpoint. Purely procedure related Serious Adverse Device Effects (SADE- $p_{Cor}$ ) are not counted.

... The primary hypothesis evaluates the SADE- $d_{Cor}$  free rate ( $Cor_{SADE\_free}$ ). It is expected, that the rate will be significantly above 90% ...

#### CIP chapter 11.1 Statistical design, method and analytical procedures

To test the primary hypothesis an exact binomial tests is carried out. Additionally, an exact 2-sided 95% confidence interval will be generated.



# 12Sec. Endpoint 1: Kaplan-Meier estimate for the Cor Family related SADE-free rate

#### 12.1 Analysis set

All analyses are performed for the Cor family analysis set<sup>105</sup> excluding the patients that are erroneously enrolled despite violation of inclusion or exclusion criteria at the time of enrollment as defined for the primary endpoint analysis.

#### 12.2 Variables

| Data file<br>record_id &<br>patient_<br>display_id_full | | | | | Nominal<br>values |
|---|---|---|---|---|---|
| event_<br>evaluation | no report | AESTDT | Onset date | date | n.a. |
| event_<br>evaluation | no report | AERELSET | Adverse Event is relevant for SADE endpoint | nominal | <ul><li>Yes</li><li>No</li></ul> |

| Data file<br>record_id &<br>patient_<br>display_id_full | Notes | | | | Nominal<br>values |
|---|---|---|---|---|---|
| data_SAR | no report | date_implantation_SAR | Date of implantation | date | n.a. |
| | no report | _ | Date of censoring (latest date of AE onset, AE resolution, implantation, PHD, 3m FU, 6m FU, 12m FU, or date of study termination) | date | n.a. |
| | no report | date_1stSADE_corfamily_SAR | Date of first Cor family related SADE | date | n.a. |
| | descriptive and<br>95% CI, Kaplan | , , _ , , _ | Any Cor family related SADE | nominal | <ul><li>Yes</li><li>No</li></ul> |
| | | | Days from implantation to first Corfamily related SADE or censoring | date | n.a. |

| _ |
|---|
| I |



See general definitions in chapter 5.4.

#### 12.4 Exclusion of Particular Information

See general definitions in chapter 5.5.

#### 12.5 Descriptive Analyses

See general definitions in chapter 5.1 and notes previous variable tables. A Kaplan-Meier survival curve has to be reported.

#### 12.6 Hypotheses & Statistical Tests

<u>CIP chapter</u> 7.2.2.1 Secondary endpoint 1: Kaplan-Meier estimate for the Cor Family related SADE-free rate

The Kaplan-Meier method will be applied to estimate the 3-month SADE-free rate at 92 days after implantation (sensitivity analysis of the primary endpoint) and the 12-month SADE-free rate at 365 days after implantation. Thereby all patients will be included in the analysis.

The pointwise 95% confidence interval has to be calculated via the loglog transformation.



### 13 Sec. Endpoint 2: Automatic LV VectorOpt test (CRT only)

#### 13.1 Analysis set

All analyses are performed for the CRT analysis set. 109

#### 13.2 Variables

CIP chapter 7.2.2.2 Secondary endpoint 2: Automatic LV VectorOpt test (CRT only)

At Pre-Hospital Discharge or at the latest at 3-month follow-up, the following endpoints related to the automatic LV VectorOpt test will be assessed:

- a. time needed to perform the LV threshold measurement manually
- b. time needed to perform the LV threshold measurement automatically
- c. investigator appraisal (score) of RV-LV conduction time test
- d. investigator appraisal (score) of intuitiveness of the threshold test
- e. investigator appraisal (score) of ease to find the best LV pacing configuration
- f. investigator appraisal (score) of overall handling of the Auto LV VectorOpt feature
- g. investigator agreement (score) to different statements relating to programmer-based LV vector optimization

| Data file identifier patient_display_id_full | | | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| auto_lv_<br>vectoropt | descriptive<br>(a) | _ | measurement manually | scale<br>hh:mm:ss has to be<br>converted to min | n.a. |
| | descriptive<br>(b)* | | measurement automatically (same subset of | scale<br>hh:mm:ss has to be<br>converted to min | n.a. |



| Data file<br>identifier<br>patient_<br>display_id_full | | Variable<br>name | Variable<br>label | level | Nominal<br>values |
|---|---|---|---|---|---|
| auto_lv_<br>vectoropt | descriptive<br>(c) | DURVLVAS<br>with "not<br>done" to be<br>analyzed as<br>missing data | time test helpful? | nominal | o No<br>o Not done |
| | descriptive<br>(d) | DUITHTAS | Intuitiveness of the threshold test | nominal | <ul><li>Very intuitive</li><li>Intuitiv</li><li>Adequate</li><li>Difficult</li><li>Very difficult</li></ul> |
| | descriptive<br>(e) | DUBLVPAS | Ease to find the best LV pacing configuration | | o Very easy o Easy o Adequate o Difficult o Very difficult |
| | descriptive<br>(f) | DULVVOAS | Overall Handling assessment of the Auto LV VectorOpt feature | nominal | o Very good o Good o Adequate o Poor o Very poor |
| | descriptive<br>(g) | DUINVAS01 | The parameters RV-LV conduction time,<br>PNS threshold and impact on device<br>longevity (pacing threshold) provide a<br>good decision basis and are sufficient for<br>a clinically acceptable LV vector<br>optimization | | <ul> <li>Strongly agree</li> <li>Somewhat agree</li> <li>Neither agree nor disagree</li> <li>Somewhat disagree</li> <li>Strongly disagree</li> </ul> |
| | descriptive<br>(g) | DUINVAS02 | Auto LV VectorOpt is an ergonomic tool<br>for informed decision making and<br>recommending which vector to select | | <ul> <li>Strongly agree</li> <li>Somewhat agree</li> <li>Neither agree nor disagree</li> <li>Somewhat disagree</li> <li>Strongly disagree</li> </ul> |
| | descriptive<br>(g) | DUINVAS03 | The automatic measurement process simplifies the process of finding a suitable LV pacing vector for CRT | nominal | <ul> <li>Strongly agree</li> <li>Somewhat agree</li> <li>Neither agree nor disagree</li> <li>Somewhat disagree</li> <li>Strongly disagree</li> </ul> |

| Data file, | Notes | Variable | Variable | Variable | nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| auto_lv_ | case listings | COITHTAS | Please specify intuitiveness of test | text | n.a. |
| vectoropt | case listings | COBLVPAS | Please specify ease of finding LV pacing configuration | text | n.a. |
| | case listings | COLVVOAS | Please specify overall assessment | text | n.a. |



See general definitions in chapter 5.4.

See time needed to perform the LV threshold measurement manually.

#### 13.4 Exclusion of Particular Information

See general definitions in chapter 5.5.

#### 13.5 Descriptive Analyses

See general definitions in chapter 5.1 and notes previous variable tables.

#### 13.6 Hypotheses & Statistical Tests

There are no pre-specified hypotheses.



### 14Sec. Endpoint 3: CRT AutoAdapt feature (CRT only)

#### 14.1 Analysis set

All analyses are performed for the CRT AutoAdapt analysis set. 110

#### 14.2 Variables

#### CIP chapter 7.2.2.2 Secondary endpoint 3: CRT AutoAdapt (CRT only)

At the 3-month follow-up the CRT AutoAdapt feature will be assessed with regard to the following endpoints:

- a. percentage of CRT pacing since last follow-up
- b. percentage of adaptive BiV pacing since last follow-up
- c. percentage of programmed BiV pacing since last follow-up
- d. percentage of adaptive LV pacing since last follow-up
- e. mean adapted AV delay after pace/sense
- f. rate of patients in whom the programming of CRT Autoadapt is maintained beyond the 3-month follow-up
- g. reasons for deactivation of CRT AutoAdapt
- h. investigator appraisal (score) of programmability
- i. investigator appraisal (score) of clinical acceptability
- j. investigator appraisal (score) of overall assessment of the CRT AutoAdapt feature

#### Lead measurements / Percentage of CRT pacing since last follow-up

The following analyses have to be performed for the data of the 3m follow-up<sup>111</sup>.

| Data file,<br>identifier<br>PRVISIT &<br>patient_<br>display_id_full | Notes | Variable<br>name | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| lead_<br>measurement | no report | PRVISIT | Visit | nominal | o 3m Follow-up |
| | descriptive (a) | DUMCRTP | Mean CRT pacing since last follow-up [%] | scale | n.a |
| | descriptive (e) | DUAVDAPO | Optimized AV delay after pace [ms] | scale | n.a. |
| | descriptive (e) | DUAVDASO | Optimized AV delay after sense [ms] | scale | n.a. |
| | 2x2 table | _ | PHD: CRT AutoAdapt "ON" M03: CRT AutoAdapt "ON" | nominal | o Yes<br>o No |



| Data file patient_display_id_full | Notes | | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| follow_up_3m | descriptive | | NEW: CRT AutoAdapt "ON" at the end of the 3mo FU | nominal | <ul><li>Yes</li><li>No</li></ul> |
| | descriptive for DUAUAON= No (g) | | Please specify why CRT AutoAdapt<br>"OFF" or "AVAdapt" | nominal | o Patient has chronic complete<br>AV block (contraindication)<br>o Other |
| | descriptive (h) | DUPRGAS | Programmability | ordinal | o Very easy o Easy o Adequate o Poor o Very poor |
| | descriptive(i) | | Clinical acceptability of the algorithm's decision | ordinal | o Very good o Good o Adequate o Poor o Very poor |
| | descriptive (j) | | Overall assessment of the<br>CRT AutoAdapt feature | ordinal | o Very good<br>o Good<br>o Adequate<br>o Poor<br>o Very poor |

| | Notes | Variable | | Variable | - |
|---|---|---|---|---|---|
| patient_ | | name | label | level | values |
| display_id_full | | | | | |
| follow_up_3m | case listings for | COAUAOTH | Other Reason for CRT AutoAdapt OFF | text | n.a. |
| | COAUAOFF = Other | | | | |
| | case listings | | Comment on programmability | text | n.a. |
| | for poor assessments | COALGRAS | comment on clinical acceptability of the | text | n.a. |
| | | | algorithm's decision | | |
| | | COAUAOAS | comment on overall assessment | text | n.a. |

#### **Home Monitoring Data**

| Data file,<br>identifier<br>date &<br>patient_<br>display_id_full | | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|---|
| _ | descriptive (b) | HMADAPBIVP | Adaptive BiV pacing since last follow-up [%] | metric | n.a. |
| (CDW<br>datamart) | descriptive (c) | HMPRGBIVP | Programmed BiV pacing since last follow-up [%] | metric | n.a. |
| | descriptive (d) | HMADAPLVP | Adaptive LV pacing since last follow-up [%] | metric | n.a. |



See general definitions in chapter 5.4.

#### 14.4 Exclusion of Particular Information

See general definitions in chapter 5.5.

#### 14.5 Descriptive Analyses

See general definitions in chapter 5.1 and notes previous variable tables.

#### 14.6 Hypotheses & Statistical Tests

There are no pre-specified hypotheses.



#### 15 Abbreviations

ADE Adverse Device Effect

AE Adverse Event
AF Atrial Fibrillation

CDMS Clinical Data Management System

CI Confidence Interval

CIP Clinical Investigation Plan

CIR Clinical Investigation Report

CRF Case listing Form

FU Follow-up

SADE Serious Adverse Device Event

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAR Statistical Analysis Report

SOP Standard Operating Procedure

SD Standard Deviation

